CLINICAL TRIAL: NCT01262976
Title: Safety and Immunogenicity of GSK Biologicals' Candidate Tuberculosis Vaccine (692342) When Administered to HIV-positive Adults Living in a Tuberculosis Endemic Region
Brief Title: Safety and Immunogenicity Study of a Candidate Tuberculosis Vaccine in Human Immunodeficiency Virus (HIV)-Positive Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 113935
Record Dates: First submitted 2010-12-16; First posted 2010-12-20 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2017-11

CONDITIONS: Tuberculosis
Keywords: Tuberculosis vaccine
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- HIV(+)-HA/GSK692342 (Experimental): HIV-infected subjects between and including 18 to 59 years of age, who were on Highly Active Anti-Retroviral Therapy (HAART) at the time of study enrolment, received two doses of GSK692342 vaccine (TB) at Day 0 and Day 30, intramuscularly into the arm's deltoid region.
  Interventions: Biological: GSK's investigational vaccine 692342
- HIV(+)-HA/Placebo (Placebo Comparator): HIV-infected subjects between and including 18 to 59 years of age, who were on Highly Active Anti-Retroviral Therapy (HAART) at the time of study enrolment, received two doses of saline solution at Day 0 and Day 30, intramuscularly into the arm's deltoid region.
  Interventions: Biological: Physiological saline
- HIV(+)-TN/GSK692342 (Experimental): HIV-infected subjects between and including 18 to 59 years of age, who were HAART-treatment naive (TN) at the time of study enrolment, received two doses of GSK692342 vaccine (TB) at Day 0 and Day 30, intramuscularly into the arm's deltoid region.
  Interventions: Biological: GSK's investigational vaccine 692342
- HIV(+)-TN/Placebo (Placebo Comparator): HIV-infected subjects between and including 18 to 59 years of age, who were HAART-treatment naive (TN) at the time of study enrolment, received two doses of saline solution at Day 0 and Day 30, intramuscularly into the arm's deltoid region.
  Interventions: Biological: Physiological saline
- HIV(-)/GSK692342 (Experimental): Subjects between and including 18 to 59 years of age, who were HIV-negative at the time of study enrolment, received two doses of GSK692342 vaccine (TB) at Day 0 and Day 30, intramuscularly into the arm's deltoid region.
  Interventions: Biological: GSK's investigational vaccine 692342
- HIV(-)/Placebo (Placebo Comparator): Subjects between and including 18 to 59 years of age, who were HIV-negative at the time of study enrolment, received two doses of saline solution at Day 0 and Day 30, intramuscularly into the arm's deltoid region.
  Interventions: Biological: Physiological saline

INTERVENTIONS:
Biological: GSK's investigational vaccine 692342 — Intramuscular, 2 doses
  Arms: HIV(+)-HA/GSK692342; HIV(+)-TN/GSK692342; HIV(-)/GSK692342
Biological: Physiological saline — Intramuscular, 2 doses
  Arms: HIV(+)-HA/Placebo; HIV(+)-TN/Placebo; HIV(-)/Placebo

SUMMARY:
The purpose of the study is to assess the safety and immunogenicity of a GlaxoSmithKline (GSK) Biologicals' candidate tuberculosis vaccine (692342) administered to Human Immunodeficiency Virus (HIV)-positive adults aged 18 to 59 years, living in a tuberculosis endemic region.

Subjects will be followed-up for 3 years.

Subjects will be enrolled in 3 cohorts:

* HIV-positive adults on highly active antiretroviral therapy
* HIV-positive adults not on highly active antiretroviral therapy
* HIV-negative adults

Each cohort will have 2 groups.

DETAILED DESCRIPTION:
This Protocol Posting has been updated following Protocol Amendment 1, February 2011, leading to the update of the outcome measures and the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* A male or female between, and including, 18 and 59 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject prior to any study procedure.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination,
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.
* Clinically acceptable laboratory values at screening as determined by the investigator.
* No evidence of tuberculosis disease with no evidence of pulmonary pathology as confirmed by chest X-ray.
* No history of extra pulmonary tuberculosis.
* Based on their medical history, all subjects must have no history of chemotherapy for tuberculosis.

Additional inclusion criteria for subjects to be enrolled in HIV+ on highly active antiretroviral therapy cohort:

* Subjects must be HIV-positive and under care of a physician for at least 6 months.
* Subjects must have a CD4+T cell count >= 250 cells/mm3 at screening.
* Subjects must be stable on highly active antiretroviral therapy for at least 6 months, with an undetectable HIV viral load level at screening.

Additional inclusion criteria for subjects to be enrolled in HIV+ treatment naïve cohort:

* Subjects must be HIV-positive and under care of a physician for at least 6 months
* Subjects must be highly active antiretroviral therapy-naïve (never received anti-retroviral therapy after HIV diagnosis)
* Subjects must have a CD4 + T cell count above 350 cells/mm3 at screening.
* Subjects for whom commencement of highly active antiretroviral therapy is not expected based on current assessment within next year.
* Subjects must have a viral load between 5000 - 80000 copies/mL at screening.

Additional inclusion criteria for subjects to be enrolled in HIV-negative cohort

• Subjects must be negative for HIV-1.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Administration of a registered live vaccine not foreseen by the study within 30 days preceding the first dose of study vaccine and administration of a registered inactivated vaccine within 14 days preceding the first dose of study vaccine.
* History of previous administration of experimental Mtb vaccines.
* History of previous exposure to components of the investigational vaccine within 30 days preceding the first dose of study vaccine
* Chronic administration of immunosuppressant or other immune-modifying drugs within six months prior to the first vaccine/product dose. For corticosteroids, this will mean prednisone >= 20 mg/kg/day, or equivalent. Inhaled and topical steroids are allowed.
* Any condition or illness or medication, which in the opinion of the Investigator might interfere with the evaluation of the safety or immunogenicity of the vaccine.
* Planned participation or participation in another experimental protocol with an experimental product during the study period.
* Administration of any immunoglobulin, any immunotherapy and/or any blood products within the three months preceding the first dose of study vaccination, or planned administrations during the study period.
* Subjects taking any of the following medication: chronic administration of systemic steroids, interleukins, systemic interferon or systemic chemotherapy.
* History of allergic reactions or anaphylaxis to any drug or vaccine.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History of chronic alcohol consumption and/or drug abuse which in the Investigator's opinion would put the subject at risk.
* Pregnant female, lactating female or female planning to become pregnant or stop contraception.
* Acute or chronic clinically relevant pulmonary, cardiovascular, hepatic or renal function abnormality as determined by physical examination or laboratory screening tests.

Additional exclusion criteria for subjects to be enrolled in HIV+ on highly active antiretroviral therapy cohort:

* Any change in anti-retroviral drug regimen within 12 weeks prior to screening.
* Any chronic drug therapy, other than highly active antiretroviral therapy or prophylaxis for opportunistic HIV related infections, birth control pills, anti-histamines for seasonal allergies and SSRIs.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2011-01-17 (Actual); Primary Completion 2012-07-17 (Actual); Study Completion 2015-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tharamani Chennai, India

REFERENCES:
- [Derived] Kumarasamy N, Poongulali S, Beulah FE, Akite EJ, Ayuk LN, Bollaerts A, Demoitie MA, Jongert E, Ofori-Anyinam O, Van Der Meeren O. Long-term safety and immunogenicity of the M72/AS01E candidate tuberculosis vaccine in HIV-positive and -negative Indian adults: Results from a phase II randomized controlled trial. Medicine (Baltimore). 2018 Nov;97(45):e13120. doi: 10.1097/MD.0000000000013120. PMID 30407329

RESULTS

PARTICIPANT FLOW:
Period: Up to Month 2
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Started | 40 | 40 | 40 | 40 | 40 | 40
Completed | 37 | 39 | 39 | 38 | 38 | 36
Not Completed | 3 | 1 | 1 | 2 | 2 | 4
Not completed — Serious Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Migrated/moved from study area | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 1 | 1
Not completed — Other | 1 | 0 | 0 | 1 | 0 | 2
Period: Up to Month 7
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Started | 40 | 40 | 40 | 40 | 40 | 40
Completed | 35 | 40 | 34 | 34 | 38 | 36
Not Completed | 5 | 0 | 6 | 6 | 2 | 4
Not completed — Serious Adverse Event | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Migrated/moved from study area | 0 | 0 | 1 | 3 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 3 | 1 | 3
Not completed — Other | 3 | 0 | 2 | 0 | 0 | 0
Period: Up to Year 1
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Started | 40 | 40 | 40 | 40 | 40 | 40
Completed | 31 | 39 | 37 | 36 | 29 | 31
Not Completed | 9 | 1 | 3 | 4 | 11 | 9
Not completed — Serious Adverse Event | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Migrated/moved from study area | 1 | 0 | 0 | 3 | 3 | 2
Not completed — Lost to Follow-up | 4 | 0 | 0 | 1 | 6 | 5
Not completed — Other | 3 | 1 | 0 | 0 | 2 | 1
Not completed — Subjects with unknown completion status | 0 | 0 | 1 | 0 | 0 | 1
Period: Up to Year 2
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Started | 40 | 40 | 40 | 40 | 40 | 40
Completed | 35 | 39 | 35 | 36 | 36 | 35
Not Completed | 5 | 1 | 5 | 4 | 4 | 5
Not completed — Serious Adverse Event | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Migrated/moved from study area | 0 | 0 | 0 | 2 | 1 | 2
Not completed — Lost to Follow-up | 1 | 1 | 2 | 2 | 3 | 3
Not completed — Subjects with unknown completion status | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 3 | 0 | 0 | 0 | 0 | 0
Period: Up to Year 3
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Started | 40 | 40 | 40 | 40 | 40 | 40
Completed | 34 | 38 | 33 | 35 | 38 | 36
Not Completed | 6 | 2 | 7 | 5 | 2 | 4
Not completed — Serious Adverse Event | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Migrated/moved from study area | 0 | 0 | 0 | 2 | 1 | 1
Not completed — Lost to Follow-up | 2 | 2 | 4 | 3 | 1 | 3
Not completed — Subjects with unknown completion status | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 3 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- HIV(+)HA-/Placebo: HIV-infected subjects between and including 18 to 59 years of age, who were on Highly Active Anti-Retroviral Therapy (HAART) at the time of study enrolment, received two doses of saline solution at Day 0 and Day 30, intramuscularly into the arm's deltoid region.
- Total: Total of all reporting groups
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)HA-/Placebo | HIV(+)-TN/GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo | Total
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40 | 240
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.0 (6.5) | 35.5 (6.2) | 32.6 (6.5) | 32.2 (5.3) | 33.9 (7.6) | 34.6 (6.4) | 34.1 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 29 | 28 | 30 | 27 | 167
  Male | 13 | 14 | 11 | 12 | 10 | 13 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: Asian - Central/South Asian Heritage | 40 | 40 | 38 | 36 | 38 | 39 | 231
  Geographic ancestry: Asian - East Asian Heritage | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Geographic ancestry: Asian - South East Asian Heritage | 0 | 0 | 2 | 3 | 2 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain and swelling. Grade 3 pain = pain that prevented normal activity. Grade 3 swelling = swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available and who had filled in the symptom sheet.
Measure: Count of Participants; unit: Participants
Groups:
- HIV(+)-TN/ GSK692342: HIV-infected subjects between and including 18 to 59 years of age, who were HAART-treatment naive (TN) at the time of study enrolment, received two doses of GSK692342 vaccine (TB) at Day 0 and Day 30, intramuscularly into the arm's deltoid region.
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/ GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
Participants
  Grade 3 Pain, Dose 1 | 1 | 0 | 1 | 0 | 2 | 0
  Grade 3 Swelling, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 37
  Grade 3 Pain, Dose 2 | 3 | 0 | 2 | 0 | 4 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 37
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Pain, Across doses | 3 | 0 | 3 | 0 | 4 | 0
  Grade 3 Swelling, Across doses | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Subjects With Grade 3 Solicited General Symptoms
Description: Solicited general symptoms assessed were fatigue, temperature [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], gastrointestinal symptoms (gastro) [nausea, vomiting, diarrhoea and/or abdominal pain], headache, malaise and myalgia. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.5 °C.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/ GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
Participants
  Grade 3 Fatigue, Dose 1 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 Gastro, Dose 1 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 Headache, Dose 1 | 0 | 1 | 0 | 0 | 3 | 0
  Grade 3 Malaise, Dose 1 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 Myalgia, Dose 1 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 Temperature, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 37
  Grade 3 Fatigue, Dose 2 | 1 | 0 | 0 | 0 | 1 | 0
  Grade 3 Gastro, Dose 2: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 37
  Grade 3 Gastro, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 37
  Grade 3 Headache, Dose 2 | 2 | 0 | 1 | 0 | 4 | 0
  Grade 3 Malaise, Dose 2: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 37
  Grade 3 Malaise, Dose 2 | 2 | 0 | 0 | 0 | 1 | 0
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 37
  Grade 3 Myalgia, Dose 2 | 1 | 0 | 0 | 0 | 1 | 0
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 37
  Grade 3 Temperature, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Fatigue, Across doses | 1 | 0 | 0 | 0 | 1 | 0
  Grade 3 Gastro, Across doses | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 Headache, Across doses | 2 | 1 | 1 | 0 | 5 | 0
  Grade 3 Malaise, Across doses | 2 | 0 | 0 | 0 | 1 | 0
  Grade 3 Myalgia, Across doses | 1 | 0 | 0 | 0 | 1 | 0
  Grade 3 Temperature, Across doses | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Subjects With Grade 3 Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset out-side the specified period of follow-up for solicited symptoms. Grade 3 AE = an AE which prevented normal, everyday activities.
Time Frame: During the 30-day (Days 0-29) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/ GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
Participants | 26 | 27 | 35 | 33 | 13 | 13

4. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From screening up to one month post Dose 2
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/ GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
Participants | 1 | 0 | 2 | 0 | 0 | 0

5. Primary Outcome: Number of Subjects With Grade 3 and Grade 4 Haematological and Biochemical Levels
Description: Haematological and biochemical parameters assessed were haemoglobin [Hgb], white blood cells [WBC], platelets [PLA], alanine aminotransferase [ALT], aspartate aminotransferase [AST] and creatinine [CREA]. The haematology and biochemistry toxicity grading scale was based on the Guidance for Industry - Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials.
Time Frame: At Day 0
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
Participants
  Grade 3 - Hgb (Change from baseline) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - Hgb (Change from baseline) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - Hgb (Decrease) | 1 | 1 | 2 | 3 | 2 | 2
  Grade 4 - Hgb (Decrease) | 2 | 0 | 1 | 0 | 0 | 0
  Grade 3 - WBC (Increase) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - WBC (Increase) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - WBC (Decrease) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - WBC (Decrease) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - PLA | 0 | 1 | 0 | 0 | 0 | 0
  Grade 4 - PLA | 0 | 0 | 1 | 0 | 0 | 0
  Grade 3 - ALT | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - ALT | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - AST | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - AST | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - CREA | 1 | 0 | 0 | 0 | 0 | 0
  Grade 4 - CREA | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Subjects With Grade 3 and 4 Haematological and Biochemical Levels
Description: as for outcome 5
Time Frame: At Day 7
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
Participants
  Grade 3 - Hgb (Change from baseline): number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 3 - Hgb (Change from baseline) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 4 - Hgb (Change from baseline): number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 4 - Hgb (Change from baseline) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - Hgb (Decrease): number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 3 - Hgb (Decrease) | 1 | 0 | 2 | 1 | 3 | 2
  Grade 4 - Hgb (Decrease): number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 4 - Hgb (Decrease) | 2 | 0 | 1 | 1 | 0 | 0
  Grade 3 - WBC (Increase): number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 3 - WBC (Increase) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - WBC (Increase): number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 4 - WBC (Increase) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - WBC (Decrease): number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 3 - WBC (Decrease) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - WBC (Decrease): number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 4 - WBC (Decrease) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - PLA: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 3 - PLA | 0 | 1 | 0 | 0 | 0 | 0
  Grade 4 - PLA: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 4 - PLA | 0 | 0 | 1 | 0 | 0 | 0
  Grade 3 - ALT: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 3 - ALT | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - ALT: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 4 - ALT | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - AST: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 3 - AST | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - AST: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 4 - AST | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - CREA: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 3 - CREA | 1 | 0 | 0 | 0 | 0 | 0
  Grade 4 - CREA: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 4 - CREA | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Subjects With Grade 3 and Grade 4 Haematological/Biochemical Levels
Description: as for outcome 5
Time Frame: At Day 30
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/ GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
Participants
  Grade 3 - Hgb (Change from baseline): number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 3 - Hgb (Change from baseline) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 4 - Hgb (Change from baseline): number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 4 - Hgb (Change from baseline) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - Hgb (Decrease): number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 3 - Hgb (Decrease) | 2 | 0 | 3 | 2 | 1 | 2
  Grade 4 - Hgb (Decrease): number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 4 - Hgb (Decrease) | 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 - WBC (Increase): number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 3 - WBC (Increase) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - WBC (Increase): number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 4 - WBC (Increase) | 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 - WBC (Decrease): number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 3 - WBC (Decrease) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - WBC (Decrease): number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 4 - WBC (Decrease) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - PLA: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 3 - PLA | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - PLA: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 4 - PLA | 0 | 0 | 1 | 0 | 0 | 0
  Grade 3 - ALT: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 3 - ALT | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - ALT: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 4 - ALT | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - AST: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 3 - AST | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - AST: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 4 - AST | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - CREA: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 3 - CREA | 1 | 0 | 0 | 0 | 0 | 0
  Grade 4 - CREA: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 4 - CREA | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Subjects With Grade 3-4 Haematological and Biochemical Levels
Description: as for outcome 5
Time Frame: At Day 37
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/ GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
Participants
  Grade 3 - Hgb (Change from baseline): number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 3 - Hgb (Change from baseline) | 0 | 1 | 0 | 0 | 0 | 1
  Grade 4 - Hgb (Change from baseline): number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 4 - Hgb (Change from baseline) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - Hgb (Decrease): number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 3 - Hgb (Decrease) | 2 | 1 | 2 | 2 | 2 | 1
  Grade 4 - Hgb (Decrease): number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 4 - Hgb (Decrease) | 1 | 0 | 0 | 0 | 0 | 1
  Grade 3 - WBC (Increase): number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 3 - WBC (Increase) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - WBC (Increase): number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 4 - WBC (Increase) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - WBC (Decrease): number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 3 - WBC (Decrease) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - WBC (Decrease): number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 4 - WBC (Decrease) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - PLA: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 3 - PLA | 0 | 0 | 1 | 0 | 0 | 0
  Grade 4 - PLA: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 4 - PLA | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - ALT: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 3 - ALT | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - ALT: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 4 - ALT | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - AST: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 3 - AST | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - AST: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 4 - AST | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - CREA: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 3 - CREA | 1 | 0 | 0 | 0 | 0 | 0
  Grade 4 - CREA: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 4 - CREA | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Subjects With Grade 3-4 Haematological/Biochemical Levels
Description: as for outcome 5
Time Frame: At Day 60
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/ GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
Participants
  Grade 3 - Hgb (Change from baseline): number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 3 - Hgb (Change from baseline) | 1 | 1 | 1 | 1 | 0 | 0
  Grade 4 - Hgb (Change from baseline): number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 4 - Hgb (Change from baseline) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - Hgb (Decrease): number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 3 - Hgb (Decrease) | 2 | 0 | 3 | 1 | 2 | 1
  Grade 4 - Hgb (Decrease): number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 4 - Hgb (Decrease) | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 - WBC (Increase): number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 3 - WBC (Increase) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - WBC (Increase): number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 4 - WBC (Increase) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - WBC (Decrease): number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 3 - WBC (Decrease) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - WBC (Decrease): number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 4 - WBC (Decrease) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - PLA: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 3 - PLA | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 - PLA: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 4 - PLA | 0 | 0 | 1 | 0 | 0 | 0
  Grade 3 - ALT: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 3 - ALT | 1 | 0 | 0 | 0 | 0 | 0
  Grade 4 - ALT: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 4 - ALT | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - AST: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 3 - AST | 1 | 0 | 0 | 0 | 0 | 0
  Grade 4 - AST: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 4 - AST | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 - CREA: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 3 - CREA | 1 | 0 | 0 | 0 | 0 | 0
  Grade 4 - CREA: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 4 - CREA | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Anti-Mycobacterium Tuberculosis Fusion Protein (M72) Specific Antibody Concentrations
Description: Concentration of M72-specific antibodies, as measured by the enzyme-linked immunosorbent assay (ELISA), were given in ELISA units per milliliter (EU/mL) and expressed as geometric mean concentrations (GMCs).
Time Frame: At Days 0, 30, 60, 210 and at Years 1, 2 and 3
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/ GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 39 | 39 | 39 | 38 | 39 | 39
EU/mL
  Anti-M72, Day 0: number analyzed (Participants) | 39 | 39 | 39 | 37 | 39 | 39
  Anti-M72, Day 0 | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4] | 1.5 [1.3 to 1.6] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4] | 1.5 [1.4 to 1.6]
  Anti-M72, Day 30: number analyzed (Participants) | 36 | 39 | 39 | 38 | 38 | 38
  Anti-M72, Day 30 | 4.9 [3.2 to 7.5] | 1.4 [1.4 to 1.4] | 6.0 [4.0 to 9.2] | 1.4 [1.4 to 1.4] | 11.2 [7.5 to 16.7] | 1.5 [1.3 to 1.8]
  Anti-M72, Day 60: number analyzed (Participants) | 37 | 38 | 38 | 38 | 36 | 35
  Anti-M72, Day 60 | 469.3 [310.8 to 708.5] | 1.5 [1.3 to 1.6] | 249.4 [142.3 to 437.2] | 1.4 [1.4 to 1.4] | 754.5 [532.6 to 1068.9] | 1.5 [1.3 to 1.8]
  Anti-M72, Day 210: number analyzed (Participants) | 35 | 39 | 33 | 33 | 37 | 35
  Anti-M72, Day 210 | 45.5 [31.4 to 66.0] | 1.4 [1.4 to 1.4] | 17.7 [11.0 to 28.5] | 1.4 [1.4 to 1.4] | 58.3 [42.2 to 80.6] | 1.5 [1.3 to 1.7]
  Anti-M72, Year 1: number analyzed (Participants) | 31 | 38 | 36 | 36 | 28 | 31
  Anti-M72, Year 1 | 28.0 [18.8 to 41.6] | 1.4 [1.4 to 1.4] | 9.3 [6.3 to 13.8] | 1.4 [1.4 to 1.4] | 29.4 [20.7 to 41.8] | 1.5 [1.3 to 1.6]
  Anti-M72, Year 2: number analyzed (Participants) | 35 | 38 | 35 | 35 | 35 | 34
  Anti-M72, Year 2 | 19.1 [12.9 to 28.1] | 1.4 [1.4 to 1.4] | 5.4 [3.7 to 7.8] | 1.4 [1.4 to 1.4] | 23.9 [17.5 to 32.5] | 1.5 [1.3 to 1.9]
  Anti-M72, Year 3: number analyzed (Participants) | 34 | 37 | 33 | 34 | 37 | 35
  Anti-M72, Year 3 | 22.0 [15.1 to 32.1] | 1.4 [1.4 to 1.4] | 4.9 [3.4 to 7.2] | 1.4 [1.4 to 1.4] | 24.3 [18.4 to 32.1] | 1.5 [1.3 to 1.7]

11. Secondary Outcome: Number of Seroconverted Subjects for M72-specific Antibodies
Description: A seroconverted subject for M72 antibodies was defined as a seronegative subject at baseline, with the appearance of M72 antibody concentration higher than or equal to (≥) the cut-off value of 2.8 EL.U/mL post vaccination. Antibody concentrations below the cut-off value of the assay were given an arbitrary value of half the cut-off value for the purpose of GMC calculation.
Time Frame: At Days 0, 30, 60, 210 and at Years 1, 2 and 3
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/ GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 39 | 39 | 39 | 38 | 39 | 39
Participants
  Anti-M72, Day 0: number analyzed (Participants) | 39 | 39 | 39 | 37 | 39 | 39
  Anti-M72, Day 0 | 0 | 0 | 1 | 0 | 0 | 2
  Anti-M72, Day 30: number analyzed (Participants) | 36 | 39 | 39 | 38 | 38 | 38
  Anti-M72, Day 30 | 23 | 0 | 27 | 0 | 35 | 1
  Anti-M72, Day 60: number analyzed (Participants) | 37 | 38 | 38 | 38 | 36 | 35
  Anti-M72, Day 60 | 36 | 1 | 37 | 0 | 36 | 1
  Anti-M72, Day 210: number analyzed (Participants) | 35 | 39 | 33 | 33 | 37 | 35
  Anti-M72, Day 210 | 34 | 0 | 29 | 0 | 36 | 2
  Anti-M72, Year 1: number analyzed (Participants) | 31 | 39 | 36 | 36 | 28 | 31
  Anti-M72, Year 1 | 30 | 0 | 29 | 0 | 27 | 1
  Anti-M72, Year 2: number analyzed (Participants) | 35 | 38 | 35 | 35 | 35 | 34
  Anti-M72, Year 2 | 33 | 0 | 24 | 0 | 34 | 1
  Anti-M72, Year 3: number analyzed (Participants) | 34 | 37 | 33 | 34 | 37 | 35
  Anti-M72, Year 3 | 33 | 0 | 22 | 0 | 36 | 1

12. Secondary Outcome: Frequency of M72-cluster of Differentiation 4 (CD4+) T-cells Expressing at Least 2 Immune Markers
Description: Among immune markers expressed after background reduction were interleukin-2 (IL-2), interferon-gamma (IFN-γ), tumour necrosis factor-alpha (TNF-α) and cluster of differentiation 40 - ligand (CD40-L). This endpoint presents results for CD4-all doubles.
Time Frame: At Days 0, 7, 30, 37, 60, 210 and at Years 1, 2 and 3
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: T-cells/million cells
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/ GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 34 | 37 | 34 | 33 | 35 | 33
T-cells/million cells
  CD4-all doubles, Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD4-all doubles, Day 0 | 176.5 [110.0 to 306.0] | 279.5 [127.0 to 519.0] | 173.0 [63.0 to 300.5] | 145.0 [82.0 to 317.0] | 216.5 [121.0 to 381.0] | 290.0 [122.0 to 489.0]
  CD4-all doubles, Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD4-all doubles, Day 7 | 1253.0 [545.0 to 6993.0] | 278.0 [198.0 to 622.5] | 693.0 [223.0 to 2147.0] | 168.5 [89.5 to 314.5] | 2352.0 [581.0 to 5353.0] | 274.0 [93.0 to 770.0]
  CD4-all doubles, Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD4-all doubles, Day 30 | 1661.0 [992.0 to 2258.0] | 306.0 [143.0 to 621.0] | 610.0 [312.0 to 1654.0] | 163.0 [71.0 to 265.0] | 1499.0 [1021.0 to 2889.0] | 312.0 [147.0 to 524.5]
  CD4-all doubles, Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD4-all doubles, Day 37 | 9060.0 [6906.0 to 15368.0] | 210.0 [138.0 to 512.0] | 5346.5 [2033.0 to 9841.5] | 94.0 [55.0 to 243.0] | 5705.0 [4217.0 to 10980.0] | 204.5 [158.0 to 405.0]
  CD4-all doubles, Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD4-all doubles, Day 60 | 7505.0 [3151.0 to 9705.0] | 230.5 [111.0 to 410.0] | 2283.5 [1618.0 to 4368.0] | 148.5 [91.0 to 244.0] | 2913.0 [1701.5 to 4113.0] | 229.5 [149.0 to 514.0]
  CD4-all doubles, Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD4-all doubles, Day 210 | 3488.0 [2035.0 to 5140.0] | 346.0 [226.0 to 579.5] | 1084.5 [502.0 to 1777.0] | 189.0 [109.0 to 358.0] | 1630.5 [1166.0 to 2400.0] | 287.0 [140.0 to 586.0]
  CD4-all doubles,Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD4-all doubles,Year 1 | 3593.0 [2224.0 to 4827.0] | 373.0 [228.0 to 470.0] | 863.0 [431.0 to 1572.0] | 191.5 [81.5 to 328.0] | 1181.0 [885.0 to 1943.0] | 274.0 [141.0 to 447.5]
  CD4-all doubles,Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD4-all doubles,Year 2 | 2982.0 [1340.0 to 4801.0] | 281.0 [198.0 to 467.0] | 449.0 [204.0 to 884.0] | 141.0 [74.0 to 280.0] | 1364.0 [782.0 to 1964.0] | 261.0 [118.0 to 649.0]
  CD4-all doubles,Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD4-all doubles,Year 3 | 3533.0 [1447.5 to 4888.0] | 320.0 [219.0 to 571.0] | 491.0 [208.0 to 1052.0] | 293.0 [187.0 to 677.0] | 1617.0 [1096.0 to 2236.0] | 316.5 [184.0 to 734.0]

13. Secondary Outcome: Frequency of M72-CD4+ T-cells Expressing Any Combination of Cytokines
Description: Among cytokines expressed after background reduction were cluster of differentiation 40-ligand (CD40-L), interleukin-2 (IL-2), interferon-gamma (IFN-γ) and tumour necrosis factor-alpha (TNF-α). This endpoint presents results for the following cytokine combinations: CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-),CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+),CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-),CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+).
Time Frame: At Days 0, 7, 30, 37, 60, 210 and at Years 1, 2 and 3
Population: The analysis was performed on the ATP cohort for immunogenicity,which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Median (Inter-Quartile Range); unit: T-cells/million cells
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/ GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 34 | 37 | 34 | 33 | 35 | 33
T-cells/million cells
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 0 | 58.5 [15.0 to 132.0] | 86.5 [30.5 to 204.5] | 1.0 [1.0 to 65.5] | 23.0 [1.0 to 77.0] | 93.0 [93.0 to 257.5] | 105.0 [19.5 to 240.5]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 7 | 525.0 [153.0 to 1759.0] | 109.5 [60.0 to 210.0] | 165.0 [58.0 to 1029.0] | 1.0 [1.0 to 71.5] | 257.5 [147.0 to 2817.0] | 125.0 [21.0 to 408.0]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 30 | 307.0 [133.0 to 792.0] | 85.0 [27.0 to 186.0] | 140.0 [25.0 to 816.0] | 1.0 [1.0 to 53.0] | 369.0 [133.0 to 1139.0] | 57.5 [18.5 to 99.0]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 37 | 2229.0 [1000.0 to 3539.0] | 76.0 [32.0 to 168.0] | 1290.5 [322.0 to 2817.5] | 19.0 [1.0 to 59.0] | 1639.0 [458.0 to 2917.0] | 57.0 [22.0 to 160.0]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 60 | 1257.0 [428.0 to 2169.0] | 59.5 [17.0 to 158.0] | 616.0 [233.0 to 943.0] | 24.0 [1.0 to 86.0] | 754.0 [320.0 to 1345.5] | 54.0 [27.0 to 107.5]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 210 | 967.0 [435.0 to 1310.0] | 117.5 [44.5 to 278.0] | 380.5 [114.0 to 775.0] | 30.0 [1.0 to 83.0] | 500.0 [307.0 to 884.0] | 106.0 [44.0 to 174.0]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Year 1 | 798.0 [412.0 to 1586.0] | 102.0 [62.0 to 196.0] | 220.0 [82.0 to 536.0] | 29.0 [1.0 to 92.5] | 410.5 [230.0 to 851.0] | 128.5 [26.0 to 204.5]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Year 2 | 685.0 [285.0 to 1141.0] | 121.0 [58.0 to 283.0] | 155.0 [31.0 to 342.0] | 1.0 [1.0 to 69.0] | 435.0 [308.0 to 853.0] | 88.0 [23.0 to 278.0]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Year 3 | 1078.0 [584.5 to 1850.0] | 117.5 [75.0 to 319.0] | 158.0 [54.0 to 389.0] | 32.0 [1.0 to 159.0] | 893.0 [456.0 to 1257.0] | 139.0 [72.0 to 347.0]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 0 | 9.0 [1.0 to 65.0] | 1.5 [1.0 to 40.0] | 1.0 [1.0 to 63.0] | 1.0 [1.0 to 19.0] | 7.0 [1.0 to 37.0] | 14.0 [1.0 to 38.0]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 7 | 110.0 [48.0 to 282.0] | 21.0 [1.0 to 80.5] | 42.0 [1.0 to 226.0] | 1.0 [1.0 to 31.0] | 119.0 [30.0 to 365.0] | 5.0 [1.0 to 34.0]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 30 | 450.0 [296.0 to 698.0] | 26.0 [1.0 to 58.0] | 204.0 [70.0 to 379.0] | 16.0 [1.0 to 46.0] | 463.0 [295.0 to 295.0] | 1.5 [1.0 to 30.5]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 37 | 1975.0 [806.0 to 3245.0] | 32.0 [1.0 to 85.0] | 671.5 [383.0 to 1040.0] | 1.0 [1.0 to 21.0] | 937.0 [654.0 to 1458.0] | 2.5 [1.0 to 44.0]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 60 | 2162.0 [1039.0 to 4464.0] | 11.0 [1.0 to 59.0] | 788.5 [788.5 to 1184.0] | 1.0 [1.0 to 33.0] | 684.0 [417.5 to 1207.0] | 9.0 [1.0 to 36.5]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 210 | 1370.0 [816.0 to 2192.0] | 32.5 [1.0 to 67.5] | 305.5 [161.0 to 678.0] | 1.0 [1.0 to 40.0] | 600.5 [326.0 to 934.0] | 15.0 [1.0 to 31.0]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Year 1 | 1536.0 [749.0 to 2594.0] | 30.0 [1.0 to 70.0] | 282.0 [139.0 to 589.0] | 1.0 [1.0 to 37.0] | 411.0 [262.0 to 780.0] | 27.5 [1.0 to 55.0]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Year 2 | 1130.0 [442.0 to 1650.0] | 1.0 [1.0 to 67.0] | 117.0 [40.0 to 421.0] | 18.0 [1.0 to 43.0] | 324.0 [168.0 to 617.0] | 27.0 [1.0 to 59.0]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Year 3 | 1321.0 [462.0 to 1869.5] | 13.5 [1.0 to 43.0] | 103.0 [39.0 to 356.0] | 32.0 [1.0 to 74.0] | 315.0 [225.0 to 538.0] | 32.5 [1.0 to 71.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 0 | 1.0 [1.0 to 27.0] | 1.0 [1.0 to 20.5] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 19.0] | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 18.5]
  CD4.CD40L(+) IL2(+)+TNFa(-)+IFNg(+), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD4.CD40L(+) IL2(+)+TNFa(-)+IFNg(+), Day 7 | 74.0 [31.0 to 255.0] | 1.0 [1.0 to 23.0] | 65.0 [1.0 to 278.0] | 1.0 [1.0 to 27.0] | 148.0 [25.0 to 413.0] | 1.0 [1.0 to 37.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 30 | 63.0 [20.0 to 130.0] | 1.0 [1.0 to 25.0] | 18.0 [1.0 to 43.0] | 1.0 [1.0 to 33.0] | 60.0 [60.0 to 95.0] | 1.0 [1.0 to 25.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 37 | 816.0 [364.0 to 1459.0] | 1.0 [1.0 to 25.0] | 507.0 [214.0 to 1184.0] | 1.0 [1.0 to 15.0] | 546.0 [313.0 to 692.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 60 | 325.0 [83.0 to 599.0] | 8.0 [1.0 to 22.0] | 127.0 [67.0 to 226.0] | 1.0 [1.0 to 20.0] | 145.5 [80.5 to 219.5] | 5.5 [1.0 to 19.5]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 210 | 128.0 [26.0 to 217.0] | 17.0 [1.0 to 32.0] | 8.5 [1.0 to 53.0] | 1.0 [1.0 to 3.0] | 77.5 [29.0 to 138.0] | 1.0 [1.0 to 26.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Year 1 | 160.0 [39.0 to 212.0] | 1.0 [1.0 to 21.0] | 53.0 [1.0 to 49.0] | 1.0 [1.0 to 1.0] | 58.0 [1.0 to 100.0] | 1.0 [1.0 to 26.5]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Year 2 | 133.0 [55.0 to 230.0] | 15.0 [1.0 to 36.0] | 20.0 [1.0 to 41.0] | 1.0 [1.0 to 1.0] | 57.0 [22.0 to 132.0] | 1.0 [1.0 to 29.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Year 3 | 120.5 [33.0 to 200.5] | 1.0 [1.0 to 24.0] | 1.0 [1.0 to 59.0] | 1.0 [1.0 to 17.0] | 60.0 [29.0 to 86.0] | 14.0 [1.0 to 23.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 0 | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 33.5] | 1.0 [1.0 to 32.0] | 1.0 [1.0 to 30.0] | 1.0 [1.0 to 20.5] | 1.0 [1.0 to 27.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 7 | 94.0 [42.0 to 172.0] | 1.0 [1.0 to 26.5] | 51.0 [26.0 to 139.0] | 1.0 [1.0 to 23.5] | 101.0 [27.0 to 252.0] | 1.0 [1.0 to 14.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 30 | 351.0 [174.0 to 507.0] | 1.0 [1.0 to 23.0] | 113.0 [13.0 to 180.0] | 1.0 [1.0 to 1.0] | 234.0 [92.0 to 554.0] | 1.0 [1.0 to 16.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 37 | 2065.0 [787.0 to 3498.0] | 1.0 [1.0 to 32.0] | 180.0 [316.0 to 1545.0] | 1.0 [1.0 to 28.0] | 1145.0 [591.0 to 1699.0] | 1.0 [1.0 to 21.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 60 | 1591.0 [855.0 to 2307.0] | 1.0 [1.0 to 13.0] | 425.5 [191.0 to 779.0] | 1.0 [1.0 to 1.0] | 510.5 [285.5 to 993.0] | 1.0 [1.0 to 42.5]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 210 | 476.0 [259.0 to 970.0] | 1.0 [1.0 to 56.5] | 78.0 [6.0 to 225.0] | 1.0 [1.0 to 42.0] | 247.0 [145.0 to 381.0] | 1.0 [1.0 to 41.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Year 1 | 484.0 [309.0 to 722.0] | 1.0 [1.0 to 40.0] | 103.0 [1.0 to 198.0] | 1.0 [1.0 to 13.0] | 185.0 [58.0 to 287.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Year 2 | 526.0 [187.0 to 757.0] | 13.0 [1.0 to 45.0] | 20.5 [1.0 to 97.0] | 1.0 [1.0 to 24.0] | 182.0 [46.0 to 308.0] | 1.0 [1.0 to 17.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Year 3 | 214.0 [58.0 to 633.0] | 1.0 [1.0 to 26.0] | 28.0 [1.0 to 100.0] | 4.0 [1.0 to 48.0] | 94.0 [16.0 to 214.0] | 1.0 [1.0 to 24.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 0 | 1.0 [1.0 to 28.0] | 15.0 [1.0 to 63.5] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 12.0] | 9.5 [9.5 to 31.0] | 19.0 [1.0 to 49.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 7 | 66.0 [23.0 to 486.0] | 1.0 [1.0 to 41.5] | 28.0 [1.0 to 141.0] | 1.0 [1.0 to 26.5] | 117.0 [34.0 to 345.0] | 13.0 [1.0 to 42.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 30 | 1.0 [1.0 to 88.0] | 1.0 [1.0 to 78.0] | 1.0 [1.0 to 68.0] | 1.0 [1.0 to 13.0] | 46.0 [1.0 to 113.0] | 1.0 [1.0 to 33.5]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 37 | 391.0 [128.0 to 1004.0] | 1.0 [1.0 to 38.0] | 214.0 [58.5 to 511.5] | 1.0 [1.0 to 2.0] | 318.0 [173.0 to 578.0] | 18.0 [1.0 to 75.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 60 | 57.0 [14.0 to 186.0] | 1.0 [1.0 to 45.0] | 28.5 [1.0 to 92.0] | 1.0 [1.0 to 1.0] | 76.5 [23.0 to 180.0] | 14.5 [1.0 to 51.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 210 | 32.0 [1.0 to 83.0] | 8.5 [1.0 to 28.0] | 18.0 [1.0 to 46.0] | 1.0 [1.0 to 36.0] | 31.5 [1.0 to 71.0] | 15.0 [1.0 to 50.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Year 1 | 39.0 [1.0 to 91.0] | 18.0 [1.0 to 44.0] | 1.0 [1.0 to 30.0] | 1.0 [1.0 to 28.0] | 35.0 [15.0 to 85.0] | 1.0 [1.0 to 35.5]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Year 2 | 72.0 [1.0 to 149.0] | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 35.0] | 1.0 [1.0 to 36.0] | 29.0 [1.0 to 71.0] | 18.0 [1.0 to 45.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Year 3 | 38.5 [17.5 to 104.5] | 22.5 [1.0 to 67.0] | 1.0 [1.0 to 1.0] | 19.0 [1.0 to 81.0] | 51.0 [21.0 to 98.0] | 14.5 [1.0 to 52.0]

14. Secondary Outcome: M72-cluster of Differentiation 4 (CD4+) T-cells Frequency Expressing Any Combination of Cytokines
Description: Among cytokines expressed after background reduction were cluster of differentiation 40-ligand (CD40-L), interleukin-2 (IL-2), interferon-gamma (IFN-γ) and tumour necrosis factor-alpha (TNF-α). This endpoint presents results for the following cytokine combination: CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+),CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-),CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+),CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-)
Time Frame: At Days 0, 7, 30, 37, 60, 210 and at Years 1, 2 and 3
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: T-cells/million cells
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/ GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 34 | 37 | 34 | 33 | 35 | 33
T-cells/million cells
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 0 | 1.0 [1.0 to 25.0] | 1.0 [1.0 to 44.0] | 1.0 [1.0 to 42.0] | 1.0 [1.0 to 38.0] | 1.0 [1.0 to 20.0] | 14.5 [1.0 to 40.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 7 | 48.0 [1.0 to 134.0] | 1.0 [1.0 to 57.0] | 34.0 [1.0 to 80.0] | 1.0 [1.0 to 26.0] | 34.0 [1.0 to 113.0] | 1.0 [1.0 to 28.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 30 | 54.0 [1.0 to 125.0] | 1.0 [1.0 to 29.0] | 35.0 [1.0 to 72.0] | 1.0 [1.0 to 34.0] | 81.0 [26.0 to 136.0] | 31.5 [1.0 to 73.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 37 | 583.0 [239.0 to 1040.0] | 17.0 [1.0 to 55.0] | 211.5 [69.0 to 456.0] | 1.0 [1.0 to 21.0] | 399.0 [251.0 to 721.0] | 1.0 [1.0 to 37.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 60 | 274.0 [50.0 to 542.0] | 1.0 [1.0 to 14.0] | 30.0 [2.0 to 103.0] | 1.0 [1.0 to 30.0] | 85.5 [43.0 to 174.0] | 1.5 [1.0 to 51.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 210 | 48.0 [3.0 to 164.0] | 27.0 [1.0 to 72.5] | 16.5 [1.0 to 112.0] | 1.0 [1.0 to 82.0] | 72.0 [12.0 to 99.0] | 4.0 [1.0 to 57.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Year 1 | 61.0 [14.0 to 141.0] | 1.0 [1.0 to 85.0] | 30.0 [1.0 to 49.0] | 2.0 [1.0 to 42.5] | 43.0 [1.0 to 82.0] | 1.0 [1.0 to 29.5]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Year 2 | 84.0 [2.0 to 110.0] | 17.0 [1.0 to 56.0] | 1.0 [1.0 to 63.0] | 1.0 [1.0 to 50.0] | 40.0 [1.0 to 89.0] | 10.0 [1.0 to 39.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Year 3 | 78.0 [45.0 to 153.5] | 1.0 [1.0 to 53.0] | 25.0 [1.0 to 70.0] | 17.0 [1.0 to 133.0] | 24.0 [1.0 to 106.0] | 8.0 [1.0 to 51.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 0 | 1.0 [1.0 to 20.0] | 4.0 [1.0 to 33.0] | 1.0 [1.0 to 12.5] | 1.0 [1.0 to 32.0] | 1.5 [1.0 to 22.5] | 7.5 [1.0 to 42.5]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 7 | 117.0 [24.0 to 209.0] | 1.0 [1.0 to 39.5] | 51.0 [1.0 to 171.0] | 1.0 [1.0 to 32.0] | 84.0 [30.0 to 255.0] | 1.0 [1.0 to 16.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 30 | 21.0 [1.0 to 58.0] | 13.0 [1.0 to 33.0] | 1.0 [1.0 to 49.0] | 1.0 [1.0 to 3.0] | 22.0 [1.0 to 43.0] | 13.5 [1.0 to 29.5]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 37 | 725.0 [287.0 to 973.0] | 1.0 [1.0 to 16.0] | 388.0 [167.5 to 694.0] | 1.0 [1.0 to 16.0] | 740.0 [399.0 to 1129.0] | 8.0 [1.0 to 24.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 60 | 74.0 [15.0 to 119.0] | 1.0 [1.0 to 23.0] | 28.5 [1.0 to 44.0] | 1.0 [1.0 to 27.0] | 55.0 [19.5 to 100.0] | 13.5 [1.0 to 45.5]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 210 | 26.0 [1.0 to 54.0] | 1.0 [1.0 to 19.0] | 1.0 [1.0 to 22.0] | 1.0 [1.0 to 17.0] | 7.5 [1.0 to 29.0] | 1.0 [1.0 to 18.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Year 1 | 15.0 [1.0 to 46.0] | 1.0 [1.0 to 18.0] | 1.0 [1.0 to 22.0] | 1.0 [1.0 to 11.5] | 13.5 [1.0 to 28.0] | 1.0 [1.0 to 14.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Year 2 | 14.0 [1.0 to 44.0] | 1.0 [1.0 to 18.0] | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 1.0] | 15.0 [1.0 to 31.0] | 1.0 [1.0 to 30.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Year 3 | 12.0 [1.0 to 46.5] | 1.0 [1.0 to 27.0] | 1.0 [1.0 to 25.0] | 1.0 [1.0 to 30.0] | 15.0 [1.0 to 43.0] | 1.0 [1.0 to 24.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 7 | 1.0 [1.0 to 150.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 30 | 1.0 [1.0 to 100.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 60.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 270.0] | 1.0 [1.0 to 170.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 37 | 1510.0 [510.0 to 3520.0] | 1.0 [1.0 to 1.0] | 300.0 [1.0 to 1170.0] | 1.0 [1.0 to 1.0] | 1400.0 [300.0 to 2330.0] | 1.0 [1.0 to 40.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 60 | 1.0 [1.0 to 1110.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 150.0] | 1.0 [1.0 to 20.0] | 1.0 [1.0 to 45.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 210 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 5.5] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Year 2 | 1.0 [1.0 to 58.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 40.0] | 1.0 [1.0 to 72.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Year 3 | 70.0 [1.0 to 835.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 360.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 230.0] | 1.0 [1.0 to 490.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 17.5] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 26.5] | 7.0 [1.0 to 38.5]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 7 | 1.0 [1.0 to 176.0] | 1.0 [1.0 to 1.0] | 21.0 [1.0 to 119.0] | 1.0 [1.0 to 1.0] | 110.0 [1.0 to 245.0] | 1.0 [1.0 to 21.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 30 | 1.0 [1.0 to 31.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 47.0] | 1.0 [1.0 to 1.0] | 26.0 [16.0 to 86.0] | 1.0 [1.0 to 23.5]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 37 | 38.0 [1.0 to 182.0] | 1.0 [1.0 to 15.0] | 123.0 [39.0 to 288.0] | 1.0 [1.0 to 1.0] | 97.0 [29.0 to 237.0] | 3.0 [1.0 to 20.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 60 | 2.0 [1.0 to 39.0] | 1.0 [1.0 to 1.0] | 40.5 [1.0 to 96.0] | 1.0 [1.0 to 1.0] | 29.0 [12.5 to 45.5] | 1.0 [1.0 to 28.5]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 210 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Year 1 | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 16.5]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Year 2 | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 29.0] | 1.0 [1.0 to 16.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Year 3 | 1.0 [1.0 to 21.5] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 21.0] | 1.0 [1.0 to 17.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 13.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 7 | 1.0 [1.0 to 18.0] | 1.0 [1.0 to 7.5] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 9.0] | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 30 | 1.0 [1.0 to 29.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 44.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 21.0] | 1.0 [1.0 to 11.5]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 37 | 43.0 [1.0 to 92.0] | 1.0 [1.0 to 1.0] | 36.5 [1.0 to 99.5] | 1.0 [1.0 to 1.0] | 19.0 [1.0 to 102.0] | 1.0 [1.0 to 14.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 60 | 26.0 [1.0 to 71.0] | 1.0 [1.0 to 1.0] | 37.5 [1.0 to 86.0] | 1.0 [1.0 to 1.0] | 19.0 [1.0 to 47.5] | 1.0 [1.0 to 15.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 210 | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Year 1 | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 20.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 9.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Year 2 | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Year 3 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 3.0]

15. Secondary Outcome: M72-CD4+ T-cells Frequency Expressing Any Combination of Cytokines
Description: Among cytokines expressed after background reduction were cluster of differentiation 40-ligand (CD40-L), interleukin-2 (IL-2), interferon-gamma (IFN-γ) and tumour necrosis factor-alpha (TNF-α). This endpoint presents results for the following cytokine combination: CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-),CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+),CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+).
Time Frame: At Days 0, 7, 30, 37, 60, 210 and at Years 1, 2 and 3
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: T-cells/million cells
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/ GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 34 | 37 | 34 | 33 | 35 | 33
T-cells/million cells
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 7 | 1.0 [1.0 to 39.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 33.0] | 1.0 [1.0 to 1.0] | 16.0 [1.0 to 56.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 19.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 37 | 46.0 [1.0 to 112.0] | 1.0 [1.0 to 1.0] | 82.0 [32.0 to 177.0] | 1.0 [1.0 to 1.0] | 36.0 [14.0 to 78.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 60 | 1.0 [1.0 to 24.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 23.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 13.5] | 1.0 [1.0 to 1.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 210 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Year 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Year 3 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 0 | 1.0 [1.0 to 27.0] | 1.0 [1.0 to 28.0] | 7.5 [1.0 to 43.0] | 17.0 [1.0 to 53.0] | 1.0 [1.0 to 42.5] | 7.0 [1.0 to 33.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 7 | 21.0 [1.0 to 90.0] | 11.0 [1.0 to 62.0] | 1.0 [1.0 to 42.0] | 1.0 [1.0 to 38.0] | 3.0 [1.0 to 48.0] | 1.0 [1.0 to 19.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 30 | 17.0 [1.0 to 57.0] | 1.0 [1.0 to 49.0] | 2.0 [1.0 to 48.0] | 9.0 [1.0 to 55.0] | 20.0 [1.0 to 80.0] | 23.0 [1.0 to 60.5]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 37 | 64.0 [1.0 to 151.0] | 1.0 [1.0 to 67.0] | 74.5 [1.0 to 190.5] | 1.0 [1.0 to 25.0] | 60.0 [6.0 to 128.0] | 1.0 [1.0 to 34.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 60 | 59.0 [5.0 to 104.0] | 21.5 [1.0 to 89.0] | 25.5 [1.0 to 84.0] | 7.5 [1.0 to 61.0] | 22.0 [1.0 to 73.0] | 1.0 [1.0 to 11.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 210 | 14.0 [1.0 to 39.0] | 1.0 [1.0 to 18.5] | 1.0 [1.0 to 21.0] | 1.0 [1.0 to 27.0] | 1.0 [1.0 to 20.0] | 1.0 [1.0 to 22.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Year 1 | 1.0 [1.0 to 30.0] | 1.0 [1.0 to 18.0] | 13.0 [1.0 to 29.0] | 1.0 [1.0 to 41.5] | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 16.5]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Year 2 | 14.0 [1.0 to 34.0] | 1.0 [1.0 to 29.0] | 1.0 [1.0 to 34.0] | 1.0 [1.0 to 58.0] | 1.0 [1.0 to 20.0] | 14.0 [1.0 to 31.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Year 3 | 1.0 [1.0 to 151.0] | 28.5 [1.0 to 189.0] | 1.0 [1.0 to 1.0] | 49.0 [1.0 to 166.0] | 21.0 [1.0 to 100.0] | 14.5 [1.0 to 132.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 0 | 1.0 [1.0 to 27.0] | 1.0 [1.0 to 39.5] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 35.0] | 1.5 [1.0 to 22.0] | 6.0 [1.0 to 30.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 7 | 29.0 [1.0 to 153.0] | 18.0 [1.0 to 62.5] | 28.0 [1.0 to 155.0] | 18.0 [1.0 to 37.0] | 68.0 [16.0 to 146.0] | 11.0 [1.0 to 33.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 30 | 1.0 [1.0 to 75.0] | 13.0 [1.0 to 60.0] | 18.0 [1.0 to 42.0] | 1.0 [1.0 to 35.0] | 17.0 [1.0 to 82.0] | 1.0 [1.0 to 53.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 37 | 85.0 [1.0 to 219.0] | 1.0 [1.0 to 22.0] | 80.5 [11.0 to 185.0] | 1.0 [1.0 to 1.0] | 56.0 [22.0 to 131.0] | 16.0 [1.0 to 51.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 60 | 18.0 [1.0 to 53.0] | 18.0 [1.0 to 51.0] | 1.0 [1.0 to 76.0] | 1.0 [1.0 to 11.0] | 29.5 [1.0 to 42.0] | 1.0 [1.0 to 29.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 210 | 1.0 [1.0 to 40.0] | 1.0 [1.0 to 51.5] | 1.0 [1.0 to 40.0] | 1.0 [1.0 to 45.0] | 1.0 [1.0 to 20.0] | 1.0 [1.0 to 30.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Year 1 | 1.0 [1.0 to 30.0] | 1.0 [1.0 to 47.0] | 6.0 [1.0 to 38.0] | 1.0 [1.0 to 42.0] | 1.0 [1.0 to 25.0] | 1.0 [1.0 to 30.5]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Year 2 | 15.0 [1.0 to 43.0] | 1.0 [1.0 to 20.0] | 1.0 [1.0 to 24.0] | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 30.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Year 3 | 8.0 [1.0 to 74.0] | 1.0 [1.0 to 43.0] | 1.0 [1.0 to 32.0] | 30.0 [1.0 to 72.0] | 1.0 [1.0 to 23.0] | 1.0 [1.0 to 24.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 0 | 5.5 [1.0 to 240.0] | 1.0 [1.0 to 311.5] | 1.0 [1.0 to 118.5] | 1.0 [1.0 to 30.0] | 1.0 [1.0 to 11.0] | 1.0 [1.0 to 198.5]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 7 | 1.0 [1.0 to 270.0] | 1.0 [1.0 to 195.0] | 1.0 [1.0 to 137.0] | 1.0 [1.0 to 150.0] | 1.0 [1.0 to 71.0] | 1.0 [1.0 to 93.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 30 | 1.0 [1.0 to 590.0] | 1.0 [1.0 to 200.0] | 40.0 [1.0 to 261.0] | 1.0 [1.0 to 150.0] | 48.0 [1.0 to 235.0] | 1.0 [1.0 to 123.5]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 37 | 120.0 [1.0 to 423.0] | 1.0 [1.0 to 104.0] | 3.5 [1.0 to 248.5] | 1.0 [1.0 to 36.0] | 320.0 [1.0 to 520.0] | 1.0 [1.0 to 150.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 60 | 1.0 [1.0 to 374.0] | 1.0 [1.0 to 97.0] | 25.5 [1.0 to 228.0] | 1.0 [1.0 to 123.0] | 1.0 [1.0 to 110.5] | 1.0 [1.0 to 166.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 210 | 32.0 [1.0 to 192.0] | 118.5 [1.0 to 276.5] | 1.0 [1.0 to 111.0] | 1.0 [1.0 to 196.0] | 37.5 [1.0 to 188.0] | 1.0 [1.0 to 167.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Year 1 | 10.0 [1.0 to 153.0] | 1.0 [1.0 to 140.0] | 7.0 [1.0 to 188.0] | 62.0 [1.0 to 204.5] | 1.0 [1.0 to 95.0] | 62.0 [1.0 to 186.5]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Year 2 | 45.0 [1.0 to 100.0] | 9.0 [1.0 to 67.0] | 1.0 [1.0 to 71.0] | 1.0 [1.0 to 46.0] | 1.0 [1.0 to 26.0] | 1.0 [1.0 to 66.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Year 3 | 8.5 [1.0 to 64.5] | 20.0 [1.0 to 102.0] | 18.0 [1.0 to 80.0] | 44.0 [1.0 to 119.0] | 1.0 [1.0 to 60.0] | 1.0 [1.0 to 96.0]
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 0 | 23.0 [1.0 to 97.0] | 2.5 [1.0 to 124.0] | 19.0 [1.0 to 98.0] | 39.0 [1.0 to 85.0] | 36.0 [1.0 to 79.0] | 34.0 [1.0 to 98.0]
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 7 | 61.0 [1.0 to 175.0] | 51.5 [1.0 to 97.5] | 15.0 [1.0 to 222.0] | 16.5 [1.0 to 110.5] | 93.0 [58.0 to 188.0] | 18.0 [1.0 to 55.0]
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 30 | 61.0 [2.0 to 104.0] | 2.0 [1.0 to 59.0] | 1.0 [1.0 to 44.0] | 40.0 [1.0 to 112.0] | 35.0 [1.0 to 72.0] | 12.5 [1.0 to 76.5]
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 37 | 135.0 [77.0 to 352.0] | 30.0 [1.0 to 79.0] | 260.0 [116.5 to 471.5] | 1.0 [1.0 to 60.0] | 245.0 [69.0 to 416.0] | 16.0 [1.0 to 63.0]
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 60 | 2.0 [1.0 to 50.0] | 17.0 [1.0 to 102.0] | 1.0 [1.0 to 35.0] | 1.0 [1.0 to 36.0] | 34.0 [4.0 to 79.5] | 25.0 [1.0 to 68.5]
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 210 | 27.0 [1.0 to 61.0] | 16.5 [1.0 to 47.5] | 12.5 [1.0 to 62.0] | 3.0 [1.0 to 37.0] | 2.5 [1.0 to 26.0] | 2.0 [1.0 to 45.0]
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Year 1 | 1.0 [1.0 to 58.0] | 1.0 [1.0 to 24.0] | 1.0 [1.0 to 30.0] | 1.0 [1.0 to 35.5] | 7.5 [1.0 to 26.0] | 12.5 [1.0 to 40.5]
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Year 2 | 1.0 [1.0 to 42.0] | 1.0 [1.0 to 22.0] | 18.0 [1.0 to 54.0] | 1.0 [1.0 to 35.0] | 1.0 [1.0 to 51.0] | 1.0 [1.0 to 30.0]
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Year 3 | 16.5 [1.0 to 53.0] | 11.0 [1.0 to 51.0] | 31.0 [1.0 to 97.0] | 45.0 [1.0 to 121.0] | 14.0 [1.0 to 57.0] | 25.0 [1.0 to 44.0]

16. Secondary Outcome: Frequency of M72-cluster of Differentiation 8 (CD8+) T-cells Expressing at Least 2 Immune Markers
Description: Among immune markers expressed after background reduction were interleukin-2 (IL-2), interferon-gamma (IFN-γ) and tumour necrosis factor-alpha (TNF-α). This endpoint presents results for CD8-all doubles.
Time Frame: At Days 0, 7, 30, 37, 60, 210 and at Years 1, 2 and 3
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: T-cells/million cells
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/ GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 34 | 37 | 34 | 33 | 35 | 33
T-cells/million cells
  CD8-all doubles, Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD8-all doubles, Day 0 | 71.5 [23.0 to 162.0] | 68.5 [31.5 to 182.5] | 58.5 [20.0 to 195.0] | 37.0 [25.0 to 164.0] | 65.0 [31.0 to 115.5] | 84.5 [36.5 to 338.5]
  CD8-all doubles, Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD8-all doubles, Day 7 | 224.0 [65.0 to 651.0] | 107.0 [46.0 to 303.5] | 149.0 [49.0 to 486.0] | 71.0 [11.0 to 229.0] | 158.0 [57.0 to 518.0] | 72.0 [39.0 to 241.0]
  CD8-all doubles, Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD8-all doubles, Day 30 | 90.0 [41.0 to 311.0] | 85.0 [22.0 to 326.0] | 60.0 [21.0 to 153.0] | 62.0 [11.0 to 129.0] | 56.0 [30.0 to 103.0] | 83.0 [44.0 to 178.0]
  CD8-all doubles, Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD8-all doubles, Day 37 | 168.0 [92.0 to 599.0] | 45.0 [20.0 to 209.0] | 179.0 [105.5 to 564.0] | 54.0 [16.0 to 146.0] | 157.0 [97.0 to 398.0] | 78.5 [43.0 to 221.0]
  CD8-all doubles, Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD8-all doubles, Day 60 | 118.0 [41.0 to 272.0] | 72.5 [24.0 to 231.0] | 91.5 [52.0 to 224.0] | 64.5 [11.0 to 205.0] | 55.0 [11.0 to 117.5] | 135.0 [56.5 to 282.5]
  CD8-all doubles, Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD8-all doubles, Day 210 | 82.0 [37.0 to 184.0] | 28.5 [11.0 to 101.0] | 42.0 [18.0 to 197.0] | 55.0 [11.0 to 104.0] | 53.5 [11.0 to 99.0] | 32.0 [11.0 to 103.0]
  CD8-all doubles, Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD8-all doubles, Year 1 | 52.0 [30.0 to 112.0] | 49.0 [11.0 to 165.0] | 47.0 [11.0 to 160.0] | 46.5 [11.0 to 100.0] | 52.0 [11.0 to 115.0] | 58.0 [11.0 to 121.0]
  CD8-all doubles, Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD8-all doubles, Year 2 | 65.0 [34.0 to 131.0] | 42.0 [20.0 to 86.0] | 46.0 [25.0 to 123.0] | 46.0 [26.0 to 90.0] | 40.0 [11.0 to 93.0] | 11.0 [11.0 to 83.0]
  CD8-all doubles, Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD8-all doubles, Year 3 | 127.5 [43.5 to 347.5] | 41.5 [17.0 to 153.0] | 48.0 [25.0 to 98.0] | 69.0 [27.0 to 120.0] | 94.0 [52.0 to 242.0] | 66.0 [42.0 to 135.0]

17. Secondary Outcome: Frequency of M72-CD8+ T-cells Expressing Any Combination of Cytokines
Description: Among cytokines expressed after background reduction were cluster of differentiation 40-ligand (CD40-L) interleukin-2 (IL-2), interferon-gamma (IFN-γ) and tumour necrosis factor-alpha (TNF-α). This endpoint presents results for the following cytokine combination: CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+),CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-),CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+),CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-),CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+).
Time Frame: At Days 0, 7, 30, 37, 60, 210 and at Years 1, 2 and 3
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: T-cells/million cells
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/ GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 34 | 37 | 34 | 33 | 35 | 33
T-cells/million cells
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 7 | 13.0 [1.0 to 143.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 55.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 110.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 37 | 1.0 [1.0 to 20.0] | 1.0 [1.0 to 1.0] | 13.0 [1.0 to 58.5] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 73.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 60 | 1.0 [1.0 to 13.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Day 210 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Year 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+), Year 3 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 21.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 7 | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 32.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 37 | 16.0 [1.0 to 33.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 21.5] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 60 | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Day 210 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Year 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-), Year 3 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+) IL2(+)+TNFa(-)+IFNg(+), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD8.CD40L(+) IL2(+)+TNFa(-)+IFNg(+), Day 7 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 11.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 39.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 37 | 1.0 [1.0 to 19.0] | 1.0 [1.0 to 1.0] | 6.0 [1.0 to 23.5] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 38.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 60 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Day 210 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Year 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+), Year 3 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 0: number analyzed (Participants) | 34 | 37 | 32 | 31 | 32 | 28
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 7 | 1.0 [1.0 to 18.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 37.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 37 | 1.0 [1.0 to 26.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 18.5] | 1.0 [1.0 to 1.0] | 26.0 [1.0 to 45.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 60 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Day 210 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Year 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-), Year 3 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 0: number analyzed (Participants) | 34 | 37 | 32 | 31 | 32 | 28
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 7 | 14.0 [1.0 to 61.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 39.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 77.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 37 | 1.0 [1.0 to 19.0] | 1.0 [1.0 to 1.0] | 6.0 [1.0 to 39.5] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 34.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 60 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Day 210 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Year 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+), Year 3 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

18. Secondary Outcome: M72-cluster of Differentiation 8 (CD8+) T Frequency Cells Expressing Any Combination of Cytokines
Description: Among cytokines expressed after background reduction were cluster of differentiation 40-ligand (CD40-L) interleukin-2 (IL-2), interferon-gamma (IFN-γ) and tumour necrosis factor-alpha (TNF-α). This endpoint presents results for the following cytokine combination: CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-),CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+),CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-),CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+),CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-).
Time Frame: At Days 0, 7, 30, 37, 60, 210 and at Years 1, 2 and 3
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: T-cells/million cells
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/ GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 34 | 37 | 34 | 33 | 35 | 33
T-cells/million cells
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 0: number analyzed (Participants) | 34 | 37 | 32 | 31 | 32 | 28
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 7 | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 37 | 1.0 [1.0 to 25.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 30.5] | 1.0 [1.0 to 1.0] | 2.0 [1.0 to 63.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 60 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Day 210 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Year 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-), Year 3 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 0 | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 7 | 1.0 [1.0 to 32.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 11.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 62.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 30 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 37 | 2.0 [1.0 to 29.0] | 1.0 [1.0 to 1.0] | 20.0 [1.0 to 49.0] | 1.0 [1.0 to 1.0] | 2.0 [1.0 to 89.0] | 1.0 [1.0 to 2.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 60 | 1.0 [1.0 to 13.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 17.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 11.5]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Day 210 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Year 1 | 1.0 [1.0 to 19.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 14.5] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Year 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+), Year 3 | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 17.0] | 1.0 [1.0 to 32.0] | 1.0 [1.0 to 20.0] | 1.0 [1.0 to 24.0] | 1.0 [1.0 to 36.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 0 | 1.0 [1.0 to 175.0] | 64.5 [1.0 to 199.5] | 155.0 [1.0 to 310.0] | 70.0 [1.0 to 220.0] | 22.0 [1.0 to 211.0] | 1.0 [1.0 to 169.5]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 7 | 72.0 [1.0 to 235.0] | 25.0 [1.0 to 168.0] | 3.0 [1.0 to 183.0] | 72.0 [1.0 to 218.0] | 74.0 [1.0 to 306.0] | 1.0 [1.0 to 150.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 30 | 1.0 [1.0 to 180.0] | 1.0 [1.0 to 130.0] | 1.0 [1.0 to 112.0] | 47.0 [1.0 to 158.0] | 210.0 [1.0 to 291.0] | 5.5 [1.0 to 128.5]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 37 | 146.0 [1.0 to 291.0] | 110.0 [1.0 to 216.0] | 23.0 [1.0 to 252.0] | 20.0 [1.0 to 83.0] | 1.0 [1.0 to 274.0] | 93.0 [1.0 to 272.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 60 | 1.0 [1.0 to 139.0] | 4.0 [1.0 to 128.0] | 1.0 [1.0 to 130.0] | 66.0 [1.0 to 190.0] | 88.5 [1.0 to 223.0] | 1.0 [1.0 to 177.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-), Day 210 | 20.0 [1.0 to 90.0] | 4.0 [1.0 to 77.5] | 1.0 [1.0 to 124.0] | 1.0 [1.0 to 52.0] | 1.0 [1.0 to 141.0] | 1.0 [1.0 to 34.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-),Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-),Year 1 | 1.0 [1.0 to 57.0] | 1.0 [1.0 to 94.0] | 1.0 [1.0 to 67.0] | 33.5 [1.0 to 132.5] | 1.0 [1.0 to 44.0] | 1.0 [1.0 to 156.5]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-),Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-),Year 2 | 1.0 [1.0 to 42.0] | 1.0 [1.0 to 47.0] | 1.0 [1.0 to 24.0] | 1.0 [1.0 to 90.0] | 18.0 [1.0 to 215.0] | 15.0 [1.0 to 183.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-),Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-),Year 3 | 1.0 [1.0 to 82.0] | 1.0 [1.0 to 10.0] | 1.0 [1.0 to 20.0] | 1.0 [1.0 to 130.0] | 1.0 [1.0 to 178.0] | 1.0 [1.0 to 109.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 11.5]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 7 | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 25.0] | 1.0 [1.0 to 26.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 17.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 30 | 1.0 [1.0 to 22.0] | 1.0 [1.0 to 12.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 37 | 1.0 [1.0 to 28.0] | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 23.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 22.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 60 | 1.0 [1.0 to 13.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 17.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Day 210 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 11.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Year 2 | 1.0 [1.0 to 12.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+), Year 3 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 7 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 30 | 1.0 [1.0 to 13.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 60: number analyzed (Participants) | 23 | 26 | 32 | 33 | 21 | 22
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 60 | 1.0 [1.0 to 13.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 37: number analyzed (Participants) | 27 | 31 | 26 | 30 | 32 | 28
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 37 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Day 210 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Year 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-), Year 3 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

19. Secondary Outcome: M72-CD8+ T-cells Frequency Expressing Any Combination of Cytokines
Description: Among cytokines expressed after background reduction were cluster of differentiation 40-ligand (CD40-L) interleukin-2 (IL-2), interferon-gamma (IFN-γ) and tumour necrosis factor-alpha (TNF-α). This endpoint presents results for the following cytokine combination: CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-),CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-),CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+).
Time Frame: At Days 0, 7, 30, 37, 60, 210 and at Years 1, 2 and 3
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: T-cells/million cells
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 34 | 37 | 34 | 33 | 35 | 33
T-cells/million cells
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 0 | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 8.5] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 7 | 1.0 [1.0 to 14.0] | 1.0 [1.0 to 12.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 30 | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 9.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 37 | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 11.0] | 1.0 [1.0 to 13.5] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 18.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 60 | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 20.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Day 210 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Year 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 12.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+), Year 3 | 1.0 [1.0 to 20.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 0 | 3.5 [1.0 to 59.0] | 1.0 [1.0 to 62.5] | 1.0 [1.0 to 5.5] | 1.0 [1.0 to 32.0] | 28.5 [1.0 to 127.5] | 1.0 [1.0 to 50.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 7 | 1.0 [1.0 to 64.0] | 17.5 [1.0 to 64.5] | 41.0 [1.0 to 87.0] | 10.5 [1.0 to 66.5] | 56.0 [1.0 to 105.0] | 1.0 [1.0 to 65.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 30 | 52.0 [1.0 to 162.0] | 1.0 [1.0 to 66.0] | 13.0 [1.0 to 46.0] | 1.0 [1.0 to 85.0] | 1.0 [1.0 to 128.0] | 5.0 [1.0 to 106.5]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 37 | 1.0 [1.0 to 84.0] | 1.0 [1.0 to 67.0] | 1.0 [1.0 to 65.0] | 1.0 [1.0 to 76.0] | 31.0 [1.0 to 163.0] | 1.0 [1.0 to 23.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 60 | 1.0 [1.0 to 49.0] | 1.0 [1.0 to 56.0] | 1.0 [1.0 to 49.0] | 1.0 [1.0 to 80.0] | 1.0 [1.0 to 59.5] | 1.0 [1.0 to 64.5]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Day 210 | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 26.5] | 10.5 [1.0 to 53.0] | 1.0 [1.0 to 46.0] | 59.5 [1.0 to 106.0] | 18.0 [1.0 to 75.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Year 1 | 1.0 [1.0 to 21.0] | 1.0 [1.0 to 55.0] | 1.0 [1.0 to 50.0] | 1.0 [1.0 to 28.0] | 1.0 [1.0 to 82.0] | 1.0 [1.0 to 28.5]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Year 2 | 1.0 [1.0 to 7.0] | 3.0 [1.0 to 52.0] | 7.5 [1.0 to 85.0] | 1.0 [1.0 to 26.0] | 1.0 [1.0 to 63.0] | 22.0 [1.0 to 76.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-), Year 3 | 1.0 [1.0 to 56.0] | 16.0 [1.0 to 136.0] | 1.0 [1.0 to 140.0] | 95.0 [1.0 to 209.0] | 1.0 [1.0 to 315.0] | 1.0 [1.0 to 92.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 0 | 35.5 [1.0 to 135.0] | 34.0 [1.0 to 90.5] | 33.0 [1.0 to 137.5] | 21.0 [1.0 to 144.0] | 9.5 [1.0 to 88.0] | 68.0 [1.0 to 316.5]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 7 | 41.0 [1.0 to 139.0] | 74.0 [1.0 to 238.5] | 27.0 [1.0 to 147.0] | 23.5 [1.0 to 135.5] | 1.0 [1.0 to 54.0] | 35.0 [1.0 to 168.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 30 | 40.0 [1.0 to 161.0] | 26.0 [1.0 to 189.0] | 9.0 [1.0 to 127.0] | 27.0 [1.0 to 86.0] | 1.0 [1.0 to 29.0] | 52.0 [1.0 to 148.5]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 37 | 59.0 [1.0 to 167.0] | 18.0 [1.0 to 157.0] | 62.5 [9.0 to 124.5] | 24.0 [1.0 to 117.0] | 23.0 [1.0 to 48.0] | 22.5 [1.0 to 186.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 60 | 33.0 [1.0 to 181.0] | 38.0 [1.0 to 135.0] | 44.5 [1.0 to 192.0] | 32.5 [1.0 to 179.0] | 1.0 [1.0 to 11.5] | 72.0 [1.0 to 211.5]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Day 210 | 36.0 [1.0 to 127.0] | 1.0 [1.0 to 67.5] | 15.5 [1.0 to 150.0] | 8.0 [1.0 to 72.0] | 1.0 [1.0 to 53.0] | 1.0 [1.0 to 61.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Year 1 | 13.0 [1.0 to 59.0] | 31.0 [1.0 to 155.0] | 25.0 [1.0 to 150.0] | 1.0 [1.0 to 70.0] | 1.0 [1.0 to 53.0] | 1.0 [1.0 to 79.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Year 2 | 20.0 [1.0 to 84.0] | 20.0 [1.0 to 54.0] | 26.5 [1.0 to 105.0] | 19.0 [1.0 to 67.0] | 1.0 [1.0 to 53.0] | 1.0 [1.0 to 46.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+), Year 3 | 60.0 [1.0 to 209.0] | 1.0 [1.0 to 119.0] | 1.0 [1.0 to 52.0] | 11.0 [1.0 to 105.0] | 57.0 [1.0 to 145.0] | 33.0 [1.0 to 55.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 0 | 1.0 [1.0 to 123.0] | 1.0 [1.0 to 39.0] | 1.0 [1.0 to 42.5] | 1.0 [1.0 to 47.0] | 1.0 [1.0 to 52.0] | 1.0 [1.0 to 81.5]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 7 | 1.0 [1.0 to 101.0] | 27.0 [1.0 to 96.5] | 29.0 [1.0 to 150.5] | 1.0 [1.0 to 30.0] | 1.0 [1.0 to 63.0] | 1.0 [1.0 to 56.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 30 | 1.0 [1.0 to 186.0] | 1.0 [1.0 to 20.0] | 16.0 [1.0 to 97.0] | 1.0 [1.0 to 47.0] | 1.0 [1.0 to 60.0] | 17.5 [1.0 to 121.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 37 | 1.0 [1.0 to 169.0] | 1.0 [1.0 to 42.0] | 1.5 [1.0 to 92.0] | 1.0 [1.0 to 49.0] | 33.0 [1.0 to 148.0] | 19.0 [1.0 to 92.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 60 | 4.0 [1.0 to 99.0] | 1.0 [1.0 to 1.0] | 20.0 [1.0 to 69.0] | 1.0 [1.0 to 41.0] | 1.0 [1.0 to 35.5] | 16.5 [1.0 to 113.5]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Day 210 | 1.0 [1.0 to 37.0] | 1.0 [1.0 to 38.0] | 35.5 [1.0 to 118.0] | 1.0 [1.0 to 55.0] | 1.0 [1.0 to 60.0] | 28.0 [1.0 to 90.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Year 1 | 1.0 [1.0 to 71.0] | 1.0 [1.0 to 41.0] | 18.0 [1.0 to 70.0] | 1.0 [1.0 to 25.0] | 1.0 [1.0 to 54.0] | 1.0 [1.0 to 66.5]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Year 2 | 36.0 [1.0 to 111.0] | 12.0 [1.0 to 52.0] | 32.5 [1.0 to 108.0] | 1.0 [1.0 to 61.0] | 3.0 [1.0 to 55.0] | 1.0 [1.0 to 46.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-), Year 3 | 1.0 [1.0 to 157.5] | 7.5 [1.0 to 156.0] | 1.0 [1.0 to 51.0] | 1.0 [1.0 to 95.0] | 1.0 [1.0 to 79.0] | 27.5 [1.0 to 129.0]
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 0: number analyzed (Participants) | 34 | 36 | 32 | 31 | 32 | 28
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 0 | 35.5 [1.0 to 416.0] | 71.0 [1.0 to 247.0] | 47.5 [1.0 to 220.0] | 50.0 [1.0 to 175.0] | 1.0 [1.0 to 98.5] | 112.5 [1.0 to 408.0]
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 7: number analyzed (Participants) | 33 | 32 | 31 | 32 | 35 | 33
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 7 | 38.0 [1.0 to 249.0] | 108.5 [1.0 to 243.5] | 30.0 [1.0 to 200.0] | 61.0 [22.0 to 165.5] | 51.0 [1.0 to 203.0] | 128.0 [21.0 to 294.0]
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 30: number analyzed (Participants) | 31 | 37 | 31 | 33 | 21 | 20
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 30 | 67.0 [1.0 to 411.0] | 50.0 [1.0 to 317.0] | 37.0 [1.0 to 94.0] | 37.0 [1.0 to 195.0] | 8.0 [1.0 to 83.0] | 93.5 [9.5 to 286.5]
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 37: number analyzed (Participants) | 27 | 31 | 32 | 33 | 21 | 22
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 37 | 65.0 [1.0 to 369.0] | 19.0 [1.0 to 134.0] | 55.0 [7.5 to 141.5] | 24.0 [1.0 to 161.0] | 29.0 [1.0 to 116.0] | 116.0 [1.0 to 268.0]
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 60: number analyzed (Participants) | 23 | 26 | 26 | 30 | 32 | 28
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 60 | 49.0 [1.0 to 203.0] | 144.5 [1.0 to 354.0] | 58.5 [1.0 to 133.0] | 75.5 [1.0 to 207.0] | 25.5 [1.0 to 134.0] | 119.5 [1.0 to 275.0]
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 210: number analyzed (Participants) | 31 | 32 | 30 | 31 | 30 | 31
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Day 210 | 79.0 [1.0 to 246.0] | 1.0 [1.0 to 70.0] | 84.5 [1.0 to 221.0] | 1.0 [1.0 to 54.0] | 40.5 [1.0 to 142.0] | 30.0 [1.0 to 150.0]
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Year 1: number analyzed (Participants) | 29 | 35 | 31 | 32 | 26 | 28
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Year 1 | 29.0 [1.0 to 121.0] | 46.0 [1.0 to 108.0] | 33.0 [1.0 to 542.0] | 33.0 [1.0 to 117.0] | 50.0 [1.0 to 110.0] | 1.5 [1.0 to 169.0]
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Year 2: number analyzed (Participants) | 27 | 37 | 34 | 29 | 31 | 31
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Year 2 | 37.0 [1.0 to 143.0] | 43.0 [1.0 to 173.0] | 43.5 [1.0 to 218.0] | 6.0 [1.0 to 66.0] | 29.0 [1.0 to 111.0] | 3.0 [1.0 to 93.0]
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Year 3: number analyzed (Participants) | 32 | 34 | 25 | 27 | 31 | 30
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+), Year 3 | 70.5 [11.0 to 219.5] | 1.0 [1.0 to 95.0] | 73.0 [1.0 to 226.0] | 44.0 [1.0 to 162.0] | 1.0 [1.0 to 114.0] | 41.0 [1.0 to 100.0]

20. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available and who had filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
Participants
  Any Pain, Dose 1 | 12 | 7 | 6 | 3 | 8 | 3
  Any Swelling, Dose 1 | 3 | 1 | 2 | 0 | 2 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 37
  Any Pain, Dose 2 | 10 | 5 | 5 | 2 | 7 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 37
  Any Swelling, Dose 2 | 4 | 0 | 2 | 0 | 4 | 0
  Any Pain, Across doses | 14 | 7 | 8 | 3 | 9 | 3
  Any Swelling, Across doses | 5 | 1 | 4 | 0 | 4 | 0

21. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Solicited general symptoms assessed were fatigue, gastrointestinal symptoms (Gastro), headache, malaise, myalgia and temperature. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
Participants
  Any Fatigue, Dose 1 | 2 | 0 | 1 | 0 | 2 | 0
  Any Gastro, Dose 1 | 1 | 0 | 1 | 0 | 2 | 1
  Any Headache, Dose 1 | 2 | 3 | 3 | 1 | 4 | 2
  Any Malaise, Dose 1 | 2 | 1 | 1 | 0 | 2 | 0
  Any Myalgia, Dose 1 | 4 | 0 | 2 | 0 | 3 | 0
  Any Temperature, Dose 1 | 0 | 1 | 2 | 2 | 3 | 0
  Any Fatigue, Dose 2: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 37
  Any Fatigue, Dose 2 | 2 | 1 | 1 | 1 | 1 | 0
  Any Gastro, Dose 2: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 37
  Any Gastro, Dose 2 | 1 | 0 | 1 | 0 | 0 | 0
  Any Headache, Dose 2: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 37
  Any Headache, Dose 2 | 4 | 2 | 2 | 1 | 8 | 0
  Any Malaise, Dose 2: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 37
  Any Malaise, Dose 2 | 2 | 1 | 1 | 0 | 1 | 0
  Any Myalgia, Dose 2: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 37
  Any Myalgia, Dose 2 | 3 | 0 | 0 | 0 | 3 | 1
  Any Temperature, Dose 2: number analyzed (Participants) | 39 | 39 | 40 | 40 | 39 | 37
  Any Temperature, Dose 2 | 5 | 0 | 4 | 1 | 9 | 1
  Any Fatigue, Across doses | 2 | 1 | 1 | 1 | 2 | 0
  Any Gastro, Across doses | 2 | 0 | 1 | 0 | 2 | 1
  Any Headache, Across doses | 4 | 3 | 4 | 2 | 8 | 2
  Any Malaise, Across doses | 2 | 2 | 1 | 0 | 2 | 0
  Any Myalgia, Across doses | 4 | 0 | 2 | 0 | 3 | 1
  Any Temperature, Across doses | 5 | 1 | 6 | 3 | 9 | 1

22. Secondary Outcome: Number of Subjects With Any Unsolicited AEs
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 30-day (Days 0-29) post-vaccination period
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
Participants | 26 | 27 | 35 | 33 | 13 | 13

23. Secondary Outcome: Number of Subjects With SAEs
Description: as for outcome 4
Time Frame: From one month post Dose 2 up to study end (Year 3)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/ GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
Participants | 2 | 0 | 2 | 0 | 0 | 0

24. Secondary Outcome: Number of Subjects Presenting Different Grades of Haematological and Biochemical Values
Description: Biochemical and haematological parameters included haemoglobin [Hgb], white blood cells [WBC], platelets [PLA], alanine aminotransferase [ALT], aspartate aminotransferase [AST] and creatinine [CREA]. Levels assessed were - normal, grade 1, grade 2 and missing grade. The haematology and biochemistry toxicity grading scale was based on the Guidance for Industry - Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials.
Time Frame: At Days 0, 7, 30, 37 and 60
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
Participants
  Normal - Hgb (Change from baseline), Day 0 | 19 | 28 | 26 | 27 | 21 | 23
  Grade 1 - Hgb (Change from baseline), Day 0 | 21 | 11 | 14 | 12 | 19 | 17
  Grade 2 - Hgb (Change from baseline), Day 0 | 0 | 1 | 0 | 1 | 0 | 0
  Missing - Hgb (Change from baseline), Day 0 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - Hgb (Change from baseline), Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Normal - Hgb (Change from baseline), Day 7 | 20 | 24 | 26 | 25 | 17 | 21
  Grade 1 - Hgb (Change from baseline), Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 1 - Hgb (Change from baseline), Day 7 | 20 | 15 | 14 | 13 | 22 | 17
  Grade 2 - Hgb (Change from baseline), Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 2 - Hgb (Change from baseline), Day 7 | 0 | 1 | 0 | 1 | 0 | 1
  Missing - Hgb (Change from baseline), Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Missing - Hgb (Change from baseline), Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - Hgb (Change from baseline), Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Normal - Hgb (Change from baseline), Day 30 | 17 | 24 | 22 | 25 | 20 | 23
  Grade 1 - Hgb (Change from baseline), Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 1 - Hgb (Change from baseline), Day 30 | 21 | 15 | 16 | 15 | 19 | 14
  Grade 2 - Hgb (Change from baseline), Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 2 - Hgb (Change from baseline), Day 30 | 1 | 1 | 2 | 0 | 0 | 0
  Missing - Hgb (Change from baseline), Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Missing - Hgb (Change from baseline), Day 30 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - Hgb (Change from baseline), Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Normal - Hgb (Change from baseline), Day 37 | 15 | 23 | 20 | 26 | 17 | 17
  Grade 1 - Hgb (Change from baseline), Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 1 - Hgb (Change from baseline), Day 37 | 22 | 15 | 16 | 12 | 21 | 19
  Grade 2 - Hgb (Change from baseline), Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 2 - Hgb (Change from baseline), Day 37 | 1 | 0 | 3 | 1 | 1 | 0
  Missing - Hgb (Change from baseline), Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Missing - Hgb (Change from baseline), Day 37 | 0 | 0 | 0 | 1 | 0 | 0
  Normal - Hgb (Change from baseline), Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Normal - Hgb (Change from baseline), Day 60 | 21 | 26 | 26 | 26 | 19 | 18
  Grade 1 - Hgb (Change from baseline), Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 1 - Hgb (Change from baseline), Day 60 | 15 | 12 | 12 | 10 | 19 | 17
  Grade 2 - Hgb (Change from baseline), Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 2 - Hgb (Change from baseline), Day 60 | 0 | 0 | 0 | 1 | 0 | 0
  Missing - Hgb (Change from baseline), Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Missing - Hgb (Change from baseline), Day 60 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - Hgb (Decrease), Day 0 | 28 | 25 | 19 | 25 | 23 | 22
  Grade 1 - Hgb (Decrease), Day 0 | 6 | 11 | 9 | 3 | 10 | 13
  Grade 2 - Hgb (Decrease), Day 0 | 3 | 3 | 9 | 9 | 5 | 3
  Missing - Hgb (Decrease), Day 0 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - Hgb (Decrease), Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Normal - Hgb (Decrease), Day 7 | 27 | 24 | 19 | 21 | 22 | 22
  Grade 1 - Hgb (Decrease), Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 1 - Hgb (Decrease), Day 7 | 7 | 11 | 11 | 7 | 9 | 11
  Grade 2 - Hgb (Decrease), Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 2 - Hgb (Decrease), Day 7 | 3 | 5 | 7 | 9 | 5 | 5
  Missing - Hgb (Decrease), Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Missing - Hgb (Decrease), Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - Hgb (Decrease), Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Normal - Hgb (Decrease), Day 30 | 23 | 22 | 17 | 22 | 21 | 22
  Grade 1 - Hgb (Decrease), Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 1 - Hgb (Decrease), Day 30 | 9 | 15 | 10 | 7 | 10 | 12
  Grade 2 - Hgb (Decrease), Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 2 - Hgb (Decrease), Day 30 | 4 | 3 | 10 | 9 | 7 | 2
  Missing - Hgb (Decrease), Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Missing - Hgb (Decrease), Day 30 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - Hgb (Decrease), Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Normal - Hgb (Decrease), Day 37 | 22 | 24 | 16 | 17 | 20 | 21
  Grade 1 - Hgb (Decrease), Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 1 - Hgb (Decrease), Day 37 | 9 | 12 | 12 | 12 | 12 | 10
  Grade 2 - Hgb (Decrease), Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 2 - Hgb (Decrease), Day 37 | 4 | 2 | 9 | 8 | 5 | 4
  Missing - Hgb (Decrease), Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Missing - Hgb (Decrease), Day 37 | 0 | 0 | 0 | 1 | 0 | 0
  Normal - Hgb (Decrease), Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Normal - Hgb (Decrease), Day 60 | 24 | 25 | 17 | 21 | 22 | 21
  Grade 1 - Hgb (Decrease), Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 1 - Hgb (Decrease), Day 60 | 9 | 10 | 13 | 9 | 9 | 10
  Grade 2 - Hgb (Decrease), Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 2 - Hgb (Decrease), Day 60 | 2 | 4 | 6 | 7 | 5 | 2
  Missing - Hgb (Decrease), Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Missing - Hgb (Decrease), Day 60 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - WBC (Increase), Day 0 | 39 | 37 | 38 | 37 | 35 | 36
  Grade 1 - WBC (Increase), Day 0 | 1 | 3 | 2 | 3 | 4 | 4
  Grade 2 - WBC (Increase), Day 0 | 0 | 0 | 0 | 0 | 1 | 0
  Missing - WBC (Increase), Day 0 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - WBC (Increase), Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Normal - WBC (Increase), Day 7 | 38 | 38 | 38 | 37 | 36 | 37
  Grade 1 - WBC (Increase), Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 1 - WBC (Increase), Day 7 | 2 | 2 | 2 | 2 | 3 | 3
  Grade 2 - WBC (Increase), Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 2 - WBC (Increase), Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Missing - WBC (Increase), Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Missing - WBC (Increase), Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - WBC (Increase), Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Normal - WBC (Increase), Day 30 | 35 | 40 | 38 | 40 | 39 | 34
  Grade 1 - WBC (Increase), Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 1 - WBC (Increase), Day 30 | 2 | 0 | 2 | 0 | 0 | 2
  Grade 2 - WBC (Increase), Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 2 - WBC (Increase), Day 30 | 1 | 0 | 0 | 0 | 0 | 2
  Missing - WBC (Increase), Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Missing - WBC (Increase), Day 30 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - WBC (Increase), Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Normal - WBC (Increase), Day 37 | 34 | 36 | 38 | 35 | 35 | 32
  Grade 1 - WBC (Increase), Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 1 - WBC (Increase), Day 37 | 4 | 3 | 0 | 4 | 4 | 4
  Grade 2 - WBC (Increase), Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 2 - WBC (Increase), Day 37 | 0 | 0 | 1 | 0 | 0 | 1
  Missing - WBC (Increase), Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Missing - WBC (Increase), Day 37 | 0 | 0 | 0 | 1 | 0 | 0
  Normal - WBC (Increase), Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Normal - WBC (Increase), Day 60 | 34 | 38 | 37 | 35 | 34 | 29
  Grade 1 - WBC (Increase), Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 1 - WBC (Increase), Day 60 | 3 | 1 | 2 | 3 | 4 | 5
  Grade 2 - WBC (Increase), Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 2 - WBC (Increase), Day 60 | 0 | 0 | 0 | 0 | 0 | 1
  Missing - WBC (Increase), Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Missing - WBC (Increase), Day 60 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - WBC (Decrease), Day 0 | 40 | 39 | 40 | 40 | 40 | 40
  Grade 1 - WBC (Decrease), Day 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 - WBC (Decrease), Day 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing - WBC (Decrease), Day 0 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - WBC (Decrease), Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Normal - WBC (Decrease), Day 7 | 39 | 40 | 40 | 39 | 39 | 40
  Grade 1 - WBC (Decrease), Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 1 - WBC (Decrease), Day 7 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 2 - WBC (Decrease), Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 2 - WBC (Decrease), Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Missing - WBC (Decrease), Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Missing - WBC (Decrease), Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - WBC (Decrease), Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Normal - WBC (Decrease), Day 30 | 38 | 39 | 40 | 40 | 39 | 38
  Grade 1 - WBC (Decrease), Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 1 - WBC (Decrease), Day 30 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 2 - WBC (Decrease), Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 2 - WBC (Decrease), Day 30 | 0 | 0 | 0 | 0 | 0 | 0
  Missing - WBC (Decrease), Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Missing - WBC (Decrease), Day 30 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - WBC (Decrease), Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Normal - WBC (Decrease), Day 37 | 35 | 38 | 39 | 39 | 39 | 37
  Grade 1 - WBC (Decrease), Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 1 - WBC (Decrease), Day 37 | 3 | 1 | 0 | 0 | 0 | 0
  Grade 2 - WBC (Decrease), Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 2 - WBC (Decrease), Day 37 | 0 | 0 | 0 | 0 | 0 | 0
  Missing - WBC (Decrease), Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Missing - WBC (Decrease), Day 37 | 0 | 0 | 0 | 1 | 0 | 0
  Normal - WBC (Decrease), Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Normal - WBC (Decrease), Day 60 | 36 | 38 | 39 | 38 | 38 | 35
  Grade 1 - WBC (Decrease), Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 1 - WBC (Decrease), Day 60 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 2 - WBC (Decrease), Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 2 - WBC (Decrease), Day 60 | 0 | 0 | 0 | 0 | 0 | 0
  Missing - WBC (Decrease), Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Missing - WBC (Decrease), Day 60 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - PLA, Day 0 | 40 | 39 | 38 | 40 | 40 | 40
  Grade 1 - PLA, Day 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 - PLA, Day 0 | 0 | 0 | 1 | 0 | 0 | 0
  Missing - PLA, Day 0 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - PLA, Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Normal - PLA, Day 7 | 40 | 39 | 39 | 39 | 39 | 40
  Grade 1 - PLA, Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 1 - PLA, Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 - PLA, Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 2 - PLA, Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Missing - PLA, Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Missing - PLA, Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - PLA, Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Normal - PLA, Day 30 | 39 | 40 | 39 | 40 | 39 | 38
  Grade 1 - PLA, Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 1 - PLA, Day 30 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 - PLA, Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 2 - PLA, Day 30 | 0 | 0 | 0 | 0 | 0 | 0
  Missing - PLA, Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Missing - PLA, Day 30 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - PLA, Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Normal - PLA, Day 37 | 38 | 38 | 38 | 39 | 38 | 37
  Grade 1 - PLA, Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 1 - PLA, Day 37 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 - PLA, Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 2 - PLA, Day 37 | 0 | 1 | 0 | 0 | 0 | 0
  Missing - PLA Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Missing - PLA Day 37 | 0 | 0 | 0 | 1 | 0 | 0
  Normal - PLA, Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Normal - PLA, Day 60 | 37 | 38 | 38 | 38 | 38 | 35
  Grade 1 - PLA, Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 1 - PLA, Day 60 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 - PLA, Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 2 - PLA, Day 60 | 0 | 0 | 0 | 0 | 0 | 0
  Missing - PLA, Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Missing - PLA, Day 60 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - ALT, Day 0 | 33 | 34 | 38 | 35 | 38 | 37
  Grade 1 - ALT, Day 0 | 6 | 6 | 2 | 5 | 2 | 3
  Grade 2 - ALT, Day 0 | 1 | 0 | 0 | 0 | 0 | 0
  Missing - ALT, Day 0 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - ALT, Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Normal - ALT, Day 7 | 30 | 32 | 34 | 34 | 35 | 35
  Grade 1 - ALT, Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 1 - ALT, Day 7 | 9 | 7 | 6 | 5 | 4 | 5
  Grade 2 - ALT, Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 2 - ALT, Day 7 | 1 | 1 | 0 | 0 | 0 | 0
  Missing - ALT, Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Missing - ALT, Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - ALT, Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Normal - ALT, Day 30 | 30 | 34 | 35 | 36 | 36 | 35
  Grade 1 - ALT, Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 1 - ALT, Day 30 | 9 | 6 | 5 | 4 | 3 | 3
  Grade 2 - ALT, Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 2 - ALT, Day 30 | 0 | 0 | 0 | 0 | 0 | 0
  Missing - ALT, Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Missing - ALT, Day 30 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - ALT, Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Normal - ALT, Day 37 | 28 | 33 | 37 | 35 | 35 | 35
  Grade 1 - ALT, Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 1 - ALT, Day 37 | 9 | 6 | 1 | 5 | 4 | 2
  Grade 2 - ALT, Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 2 - ALT, Day 37 | 1 | 0 | 1 | 0 | 0 | 0
  Missing - ALT, Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Missing - ALT, Day 37 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - ALT, Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Normal - ALT, Day 60 | 30 | 32 | 34 | 34 | 35 | 33
  Grade 1 - ALT, Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 1 - ALT, Day 60 | 6 | 7 | 5 | 4 | 3 | 2
  Grade 2 - ALT, Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 2 - ALT, Day 60 | 0 | 0 | 0 | 0 | 0 | 0
  Missing - ALT, Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Missing - ALT, Day 60 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - AST, Day 0 | 34 | 31 | 35 | 30 | 37 | 38
  Grade 1 - AST, Day 0 | 5 | 9 | 5 | 10 | 2 | 2
  Grade 2 - AST, Day 0 | 1 | 0 | 0 | 0 | 1 | 0
  Missing - AST, Day 0 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - AST, Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Normal - AST, Day 7 | 33 | 30 | 32 | 30 | 33 | 36
  Grade 1 - AST, Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 1 - AST, Day 7 | 6 | 10 | 7 | 9 | 5 | 4
  Grade 2 - AST, Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 2 - AST, Day 7 | 1 | 0 | 1 | 0 | 1 | 0
  Missing - AST, Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Missing - AST, Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - AST, Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Normal - AST, Day 30 | 32 | 33 | 33 | 30 | 33 | 35
  Grade 1 - AST, Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 1 - AST, Day 30 | 6 | 7 | 7 | 9 | 5 | 3
  Grade 2 - AST, Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 2 - AST, Day 30 | 1 | 0 | 0 | 1 | 1 | 0
  Missing - AST, Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Missing - AST, Day 30 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - AST, Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Normal - AST, Day 37 | 29 | 32 | 30 | 29 | 35 | 36
  Grade 1 - AST, Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 1 - AST, Day 37 | 8 | 7 | 9 | 11 | 4 | 1
  Grade 2 - AST, Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 2 - AST, Day 37 | 1 | 0 | 0 | 0 | 0 | 0
  Missing - AST, Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Missing - AST, Day 37 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - AST, Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Normal - AST, Day 60 | 28 | 31 | 27 | 27 | 33 | 30
  Grade 1 - AST, Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 1 - AST, Day 60 | 8 | 7 | 12 | 11 | 4 | 5
  Grade 2 - AST, Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 2 - AST, Day 60 | 0 | 1 | 0 | 0 | 1 | 0
  Missing - AST, Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Missing - AST, Day 60 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - CREA, Day 0 | 39 | 40 | 40 | 40 | 40 | 40
  Grade 1 - CREA, Day 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 - CREA, Day 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing - CREA, Day 0 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - CREA, Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Normal - CREA, Day 7 | 39 | 40 | 40 | 39 | 38 | 40
  Grade 1 - CREA, Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 1 - CREA, Day 7 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 - CREA, Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Grade 2 - CREA, Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Missing - CREA, Day 7: number analyzed (Participants) | 40 | 40 | 40 | 39 | 39 | 40
  Missing - CREA, Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - CREA, Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Normal - CREA, Day 30 | 38 | 40 | 40 | 40 | 39 | 38
  Grade 1 - CREA, Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 1 - CREA, Day 30 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 - CREA, Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Grade 2 - CREA, Day 30 | 0 | 0 | 0 | 0 | 0 | 0
  Missing - CREA, Day 30: number analyzed (Participants) | 39 | 40 | 40 | 40 | 39 | 38
  Missing - CREA, Day 30 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - CREA, Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Normal - CREA, Day 37 | 37 | 39 | 39 | 40 | 39 | 37
  Grade 1 - CREA, Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 1 - CREA, Day 37 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 - CREA, Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Grade 2 - CREA, Day 37 | 0 | 0 | 0 | 0 | 0 | 0
  Missing - CREA, Day 37: number analyzed (Participants) | 38 | 39 | 39 | 40 | 39 | 37
  Missing - CREA, Day 37 | 0 | 0 | 0 | 0 | 0 | 0
  Normal - CREA, Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Normal - CREA, Day 60 | 36 | 39 | 39 | 38 | 38 | 35
  Grade 1 - CREA, Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 1 - CREA, Day 60 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 - CREA, Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Grade 2 - CREA, Day 60 | 0 | 0 | 0 | 0 | 0 | 0
  Missing - CREA, Day 60: number analyzed (Participants) | 37 | 39 | 39 | 38 | 38 | 35
  Missing - CREA, Day 60 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: during the 30-day (Days 0-29) post-vaccination period; SAEs: during the entire study period (from Day 0 up to Year 3).
Arm/Group | HIV(+)-HA/GSK692342 | HIV(+)-HA/Placebo | HIV(+)-TN/GSK692342 | HIV(+)-TN/Placebo | HIV(-)/GSK692342 | HIV(-)/Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 2/40 | 0/40 | 0/440 | 0/40
Serious Adverse Events (participants affected / at risk) | 2/40 | 0/40 | 3/40 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 29/40 | 29/40 | 33/40 | 33/40 | 19/40 | 13/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV(+)-HA/GSK692342 (N=40) | HIV(+)-HA/Placebo (N=40) | HIV(+)-TN/GSK692342 (N=40) | HIV(+)-TN/Placebo (N=40) | HIV(-)/GSK692342 (N=40) | HIV(-)/Placebo (N=40)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cavernous sinus thrombosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV(+)-HA/GSK692342 (N=40) | HIV(+)-HA/Placebo (N=40) | HIV(+)-TN/GSK692342 (N=40) | HIV(+)-TN/Placebo (N=40) | HIV(-)/GSK692342 (N=40) | HIV(-)/Placebo (N=40)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 3 (3) | 4 (4) | 2 (2) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (7) | 4 (5) | 1 (1) | 2 (3)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2) | 7 (7) | 5 (5) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 5 (7) | 3 (3) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 5 (6) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (5) | 2 (3) | 5 (8) | 1 (1) | 2 (3) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 9 (12) | 3 (5) | 5 (6) | 7 (7) | 9 (13) | 4 (5)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Lipoatrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (4) | 2 (2) | 1 (2) | 0 (0) | 2 (3) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (8) | 0 (0) | 3 (3) | 1 (1) | 3 (6) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (7) | 4 (4) | 6 (7) | 4 (4) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 16 (24) | 10 (15) | 10 (14) | 8 (11) | 10 (16) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6) | 4 (4) | 6 (7) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 8 (8) | 7 (9) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 6 (6) | 2 (2) | 7 (10) | 6 (6) | 9 (12) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Swelling (General disorders) | 5 (7) | 1 (1) | 4 (4) | 0 (0) | 4 (6) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.